Symphogen A/S

Sym015-01

An Open-label, Multicenter Phase 1a/2a Trial Investigating the Safety, Tolerability and Antitumor Activity of Multiple Doses of Sym015, a Monoclonal Antibody Mixture Targeting MET, in Patients with Advanced Solid Tumor Malignancies

Statistical Analysis Plan

Version: Final

Project Number: 223276

### SPONSOR SIGNATURE PAGE



14-Jun-2019

Date (DD Mmm YY)

Statistical Consultant



20-Jun-2019

Date (DD Mmm YY)

PK Specialist

Symphogen A/S Sym015-01

Statistical Analysis Plan



Signatures below confirm that the Statistical Analysis Plan was developed in accordance with SOP-GDO-WW-019 and that it is approved for release.

This document has been approved and signed electronically on the final page by the following:

| Signatory |
|----------------------------------|
| Project Role: Biostatistics Lead |

## TABLE OF CONTENTS

| 1 | INTRODUCTION | 12 |
|---|---|---|
| 2 | STUDY OBJECTIVES | 14 |
| 2.1 | Objectives of Part 1, Dose-Escalation | 14 |
| 2.1.1 | Primary Objective | 14 |
| 2.1.2 | Secondary Objective(s) | 14 |
| 2.2 | Objectives of Part 2 | 14 |
| 2.2.1 | Primary Objective | 15 |
| 2.2.2 | Secondary Objective(s) | 15 |
| 3 | INVESTIGATIONAL PLAN | 15 |
| 3.1 | Overall Study Design and Plan. | 15 |
| 3.2 | Endpoints and Associated Variables | 18 |
| 3.2.1 | Efficacy Variables | 19 |
| 3.2.1 | | 19 |
| 3.2.1 | 2 Pharmacodynamic Variables | 26 |
| 3.2.1 | 3 Immunogenicity Variables | 28 |
| 3.2.2 | Pharmacokinetic Variables | 28 |
| 3.2.3 | Safety Variables | 31 |
| 3.2.3 | | 31 |
| 3.2.3 | 2 Adverse Events (AE) Survey | 31 |
| 3.2.3 | 3 Dose-Limiting Toxicities Evaluation (Part 1 Only) | |
| 3.2.3 | | |
| 3.2.3 | | 39 |
| 3.2.3 | | .40 |
| 3.2.3 | 7 Electrocardiograms (ECG) | .40 |
| 3.2.3 | Control of the control of the contro | .40 |
| 3.2.3 | | |
| 4 | STATISTICAL METHODS | |
| 4.1 | Data Quality Assurance | .42 |
| 4.2 | General Presentation Considerations | |
| 4.2.1 | Baseline | |
| 4.2.2 | End of Treatment (EOT) | .42 |
| 4.2.3 | Unscheduled assessments | |
| 4.2.4 | Treatment Day | |
| 4.2.5 | Missing Data | |
| 4.2.6 | Data Listing | .45 |
| 4.2.7 | Tables and Descriptive Statistics | 45 |
| 4.2.8 | Figures | .47 |
| 4.3 | Software48 | |
| 4.4 | Study Patients | |
| 4.4.1 | Disposition of Patients | .48 |
| 4.4.2 | Protocol Deviations | |
| 4.5 | Analysis Sets | .49 |

| 4.6 Demographics and Baseline Characteristics, Disease History and Prior Canc | er Therapies |
|---|---|
| 4.7 Medical History | 52 |
| 4.8 Prior and Concomitant Medications and Concomitant Procedures | |
| 4.9 Pre-medications for Sym015 | |
| 4.10 Treatment Exposure and Compliance | |
| 4.11 Efficacy Evaluation | |
| 4.11.1 Analysis and Data Conventions | |
| 4.11.1.1 Multi-center Studies. | |
| 4.11.1.2 Adjustments for Covariates | 56 |
| 4.11.1.3 Handling of Dropouts or Missing Data | 56 |
| 4.11.1.4 Multiple Comparisons/Multiplicity | |
| 4.11.1.5 Interim Analyses | 56 |
| 4.11.1.6 Examination of Subgroups | |
| 4.11.2 Analysis of Efficacy Variable | |
| 4.11.2.1 Anti-Tumor Response according to RECIST v1.1 | |
| 4.11.3 Pharmacodynamic and Immunogenicity | |
| 4.11.4 Pharmacokinetics | |
| 4.11.4.1 Pharmacokinetic Concentrations | |
| 4.11.4.2 Handling of Values Below the Limit of Quantification (BLQ) | |
| 4.11.4.3 Pharmacokinetic Parameters. | |
| 4.11.4.4 Pharmacokinetic Analysis | |
| 4.12 Safety Evaluation. | |
| 4.12.1 Dose Limiting Toxicities (DLT) | |
| 4.12.2 Adverse Events | |
| 4.12.3 Deaths, Serious Adverse Events, and Other Significant Adverse Events. | |
| 4.12.4 Clinical Laboratory Evaluation. | |
| 4.12.5 Echocardiogram (ECHO) or Multi-Gated (MUGA) Scan | |
| 4.12.6 Vital Signs | |
| 4.12.7 Electrocardiograms (ECG) | |
| 4.12.8 Physical Examination | |
| 4.12.9 Eastern Cooperative of Oncology Group (ECOG) Performance Status (P | |
| 4.13 Safety Monitoring. | |
| 4.14 Other Analyses | |
| 4.15 Determination of Sample Size | |
| 4.16 Changes in the Conduct of the Study or Planned Analysis | |
| 5 REFERENCES | |
| 6 TABLES, FIGURES and LISTINGS | |
| 7 APPENDICES | |
| 7.1 Derivation of CTCAE Grade - Hematological Tests | |
| 7.2 Derivation of CTCAE Grade - Clinical Chemistry Tests | 79 |
| 7.3 Derivation of CTCAE Grade - Coagulation Tests | |
| 7.4 Schedule of Assessments – Part 1 and Part 2 Basket Cohort | |
| 7.5 Schedule of Assessments – Part 2 NSCLC Cohort | |

Symphogen A/S Sym015-01

Statistical Analysis Plan

## **REVISION HISTORY**

| Version No. | Effective Date | Summary of Change(s) |
|-------------|----------------|-----------------------------------------|
| Draft 0.1 | 25 May 2016 | New document |
| Draft 1.0 | 12 Aug 2016 | Document Review |
| Draft 2.0 | Feb 2017 | Document Review |
| Draft 0.3 | 22 Feb 2019 | Use of new template and Document Review |
| Draft 0.4 | 23 Apr 2019 | Document Review |
| Draft 0.5 | 22 May 2019 | Comment Resolution |
| 1.0 | 05 Jun 2019 | Final |

## LIST OF ABBREVIATIONS

List and define all acronyms and abbreviations used in the document here. Abbreviations should be spelled out in full and the abbreviation indicated in parentheses at first appearance in the text. Abbreviations should appear in alphabetical order.

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| 1M FUP | One-Month Follow-up |
| ADA | Anti-Drug Antibody |
| ADCC | Antibody-Dependent Cellular Cytotoxicity |
| AE | Adverse event |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| ANC | Absolute Neutrophil Count |
| ASCO | American Society of Clinical Oncology |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical therapeutic chemical |
| AUC | Area under the concentration-time curve |
| AUC τ | Area under the concentration-time curve in a dosing interval |
| AUCNorm. t | Dose-normalized area under the concentration-time curve in a dosing interval |
| BLQ | Below the lower limit of quantification |
| BMI | Body Mass Index |
| BUN | Blood Urea Nitrogen |
| C#/D# | Cycle # / Day # |
| CAP | College of American Pathologists |
| CEC | Central Ethical Committee |
| CI | Confidence Interval |
| CISH | Chromogenic In Situ Hybridization |
| CL | Clearance |
| CNS | Central Nervous System |
| Cmax | Maximum Concentration |

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Project Document Version No. 1.0 Project Document Effective Date: 05Jun2019 

Symphogen A/S Sym015-01

Statistical Analysis Plan

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| CR | Complete Response |
| CRF | Case Report Form |
| CSP | Clinical Study Protocol |
| CSR | Clinical Study Report |
| CT | Computed Tomography |
| CTAE | Common Terminology Criteria for Adverse Events |
| Ctrough | Trough Concentration |
| CV | Coefficient of variation |
| Cz | Last Quantifiable Concentration |
| DLT | Dose-Limiting Toxicity |
| DRM | Data Review Meeting |
| DSUR | Development Safety Update Report |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| EOI | End of Infusion |
| EOT | End of Treatment |
| FAS | Full Analysis Set |
| FISH | Fluorescence In Situ Hybridization |
| FUP | Follow-up |
| GCP | Good Clinical Practice |
| НА | Health Authority |
| hCG | Human Chorionic Gonadotropin |
| HGF | Hepatocyte Growth Factor |
| HIV | Human immunodeficiency virus |
| ICH | International Council for Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| IEC | Independent Ethics Committee |
| lgGl | Immunoglobulin G1 |
| TD CDO 1171/ 122 01 | |

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Project Document Version No. 1.0
Project Document Effective Date: 05Jun2019


Symphogen A/S Sym015-01

Statistical Analysis Plan

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| IHC | Immunohistochemistry |
| IMP | Investigational Medicinal Product |
| INR | International Normalized Ratio |
| IRB | Institutional Review Board |
| IRR | Infusion-Related Reaction |
| ISF | Investigator Site File |
| ΓV | Intravenous |
| KRAS | Kirsten Rat Sarcoma |
| LLN | Lower Limit of Normal |
| LLOQ | Lower limit of quantification |
| LOQ | Limit of quantification |
| mAb | Monoclonal Antibody |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MET | MET proto-oncogene, hepatocyte growth factor receptor gene |
| MET <sup>Ex14Del</sup> | MET exon 14 skipping alteration |
| MRI | Magnetic Resonance Image/Imaging |
| MTD | Maximum tolerated dose |
| MUGA | Multi-Gated Acquisition |
| NA | Not available |
| NCS | Not clinically significant |
| NE | Not Evaluable |
| NGS | Next-Generation Sequencing |
| NK | Not known |
| NOAEL | No Observed Adverse Effect Level |
| NSAID | Nonsteroidal Anti-Inflammatory Drug |
| NSCLC | Non-Small Cell Lung Cancer |
| NYHA | New York Heart Association |
| OR | Objective Response |
| OTC | Over the counter |
| PD | Progressive Disease |
| TP_CDO_WW_122_01 | COMEIDENTIAL Project December 10 |

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Project Document Effective Date: 05Jun2019


Symphogen A/S Sym015-01

Statistical Analysis Plan

| Abbreviation / Acronym | Definition / Expansion |
|---|---|
| PDX | Patient-Derived Xenograft |
| PK | Pharmacokinetic |
| PR | Partial Response |
| PS | Performance Status |
| PSA | Prostate-Specific Antigen |
| PT | Preferred Term |
| PTT | Partial Thromboplastin Time |
| Q2W | Every Second Week |
| qPCR | Quantitative PCR |
| QT | The QT interval is measured from the beginning of the QRS complex to the end of the T wave |
| QTc | corrected QT interval |
| QTcB | QT corrected using Bazzett's formula |
| QTcF | QT corrected using Fridericia's formula |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| RP2D | Recommended Phase 2 Dose |
| RTK | Receptor Tyrosine Kinase |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation or Stable Disease (meaning to be extrapolated by the context) |
| SISH | Silver In Situ Hybridization |
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |
| SOI | Start of Infusion |
| SOP | Standard Operating Procedure(s) |
| SUSAR | Suspected Unexpected Serious Adverse Reactions |
| T½ | Terminal elimination half-life |
| TEAE | Treatment-emergent adverse event |
| T <sub>max</sub> | Time of Maximum Concentration |

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Project Document Effective Date: 05Jun2019


Symphogen A/S Sym015-01

Statistical Analysis Plan

| Abbreviation / Acronym I | Definition / Expansion |
|--------------------------|------------------------|
|--------------------------|------------------------|

ULN

Upper Limit of Normal

 $V_{z}$ 

Volume of distribution during the terminal phase

WHO-DD

World Health Organisation - Drug Dictionary

WT

Wild-Type

 $\lambda_z$ 

Terminal Rate Constant

CONFIDENTIAL.


Symphogen A/S Sym015-01

Statistical Analysis Plan

1 INTRODUCTION

Cancers are malignant tumors formed by an abnormal growth of cells and tissue leading to organ

failure. They fall into two categories: solid and hematological cancers. Solid tumors are formed by

an abnormal growth of body tissue cells other than blood, bone marrow or lymphatic cells. A solid

tumor consists of an abnormal mass of cells, which may stem from different tissue types such as

lung, breast, colon, prostate, stomach and liver, and which initially grows in the organ of its cellular

origin. In advanced stages of the disease, solid tumors may spread to other organs through

metastatic tumor growth. Cancer is the second-leading cause of death and disability in the world.

Lung, breast, colorectal, prostate and stomach cancer are the most common malignancies [1]. Non-

small cell lung cancer (NSCLC) is the leading cause of death due to malignancy globally [2].

MET (MET proto-oncogene tyrosine kinase, hepatocyte growth factor receptor, also known as c-

MET) is a receptor tyrosine kinase (RTK) containing an extracellular ligand-binding domain, a

transmembrane domain, and an intracellular domain with tyrosine kinase activity. The hepatocyte

growth factor (HGF), also known as scatter factor, is the only known ligand for MET. Binding of

HGF to MET leads to receptor dimerization and autophosphorylation, which activates downstream

signaling pathways and ultimately leads to increased cell proliferation, survival, and motility.

Dysregulation of MET or HGF activity plays a role in many cancers by facilitating cancer

invasiveness, angiogenesis, metastasis, and tumor growth, thus leading to a more aggressive cancer

phenotype and a poorer prognosis.

Recent preclinical and clinical results have indicated that MET (MET proto-oncogene, hepatocyte

growth factor receptor gene)-amplification confers addiction to this receptor in cancer cells and

make them susceptible to treatment with MET-targeted therapeutics [4][5].

Sym015 is a recombinant antibody mixture containing 2 humanized IgG1 mAbs, designated

Hu9006 and Hu9338, which bind specifically to MET, the receptor for HGF. Preclinical studies

have shown that Sym015 effectively down-regulates the target and has superior tumor growth

inhibitory activity compared to other antibodies targeting this receptor. Sym015 is intended for the

treatment of solid tumor malignancies with amplification of the gene encoding MET.

Symphogen A/S Sym015-01

Statistical Analysis Plan

The investigational medicinal product (IMP) tested in this trial is Sym015. This is the first clinical trial to study Sym015.

The Statistical Analysis Plan (SAP) details the statistical methodology to be used in analyzing study data and outlines the statistical programming specifications, tables, figures, and listings. It describes the variables and populations, anticipated data transformations and manipulations, and other details of the analyses not provided in the clinical study protocol. This SAP covers the planned analysis of all data collected on paper (source documents /case report forms [CRFs]), captured electronically in Data Labs, and provided by external vendors. PKand immunogenicity blood samples are analyzed by external.

Biomarker blood samples are analyzed by external laboratory

The analyses described are based on the Clinical Study Protocol (CSP) Version 8.0 (07-Dec-2018): Sym015 (Anti-MET) in Patients with Advanced Solid Tumor Malignancies, incorporating Amendment No.6, dated 20 November 2017, Amendment No. 5, dated 11 May 2017, Amendment No.4, dated 04 November 2016, Amendment No.3, dated 02 May 2016, Amendment No.2, dated 02 Feb 2016, Amendment No.1, dated 17 December 2016, and original CSP Version Final 1.0, dated 01 December 2015.

The SAP will be finalized prior to database lock and describes the statistical analysis as it is foreseen when the study is being planned. If circumstances should arise during the study rendering this analysis inappropriate, or if in the meantime improved methods of analysis should come to light, different analyses may be made. If this occurs, the sponsor will determine how the revision impacts the study and how the SAP revision should be implemented. The details of the revision will be documented and described in the clinical study report (CSR)

The structure and content are based upon ICH requirements as detailed in ICH E3 Structure and Content of Clinical Study Reports [8].

Symphogen A/S Sym015-01

Statistical Analysis Plan

2 STUDY OBJECTIVES

2.1 Objectives of Part 1, Dose-Escalation

Part 1 is the Phase 1a dose-escalation portion of the study, conducted in patients with Kirsten Rat

Sarcoma proto-oncogene (KRAS) wild-type (WT) advanced solid tumor malignancies without

available therapeutic options.

2.1.1 Primary Objective

To assess the safety and tolerability of Sym015 when administered by IV infusion on a Every

Second Week (Q2W) schedule to patients with KRAS wild-type (WT) advanced solid tumor

malignancies without available therapeutic options.

2.1.2 Secondary Objective(s)

1. To determine a Q2W Recommended Phase 2 Dose (RP2D) of Sym015

2. To evaluate the PK profile of Sym015

3. To evaluate target-engagement in skin biopsy tissue

4. To evaluate the immunogenicity of Sym015

5. To evaluate potential pharmacodynamic biomarkers of Sym015 action, and estimate, if

feasible, the magnitude of biological activity

6. To make a preliminary evaluation of the antitumor activity of Sym015

2.2 Objectives of Part 2

Part 2 is the Phase 2a dose-expansion portion of the study in which dosing will be at the

recommended Phase 2 dose (RP2D) on a biweekly (Q2W) schedule. Three patient cohorts, as

defined later in section 3.1, will be included.

Symphogen A/S Sym015-01

Statistical Analysis Plan

2.2.1 Primary Objective

To evaluate the antitumor activity of Sym015 when administered at the Q2W RP2D to patients in

the following cohorts:

1. Basket Cohort

2. NSCLC MET-Amplified Cohort

3. NSCLC MET<sup>Ex14Del</sup> Cohort

2.2.2 Secondary Objective(s)

1. To further evaluate the safety and tolerability of Sym015 when administered at the Q2W

RP2D

2. To further evaluate the PK profile of Sym015 when administered at the Q2W RP2D

3. To further evaluate the immunogenicity of Sym015 when administered at the Q2W RP2D

4. To further evaluate potential pharmacodynamic biomarkers of Sym015 action, and

estimate, if feasible, the magnitude of biological activity when administered at the Q2W

RP2D

Above secondary efficacy objectives at points 1 to 4 will be studied in the three Part 2

cohorts. Additionally, these will also be assessed on a subset of the Basket cohort as

detailed in below point 5.

5. Basket Cohort: To make a preliminary assessment of the antitumor activity of Sym015,

and to evaluate all of the above secondary objectives, in a subset of approximately 6

patients with solid tumor malignancies administered Sym015 at the Q2W RP2D after

having received prior therapy with a MET-targeting TKI.

3 INVESTIGATIONAL PLAN

Overall Study Design and Plan

This is an open-label, multicenter trial composed of 2 parts:

Symphogen A/S Sym015-01

Statistical Analysis Plan

### **Dose-Escalation Phase**

Part 1 is the Phase 1a dose-escalation portion of the study conducted in patients with KRAS wild-type (WT) advanced solid tumor malignancies without available therapeutic options. During Part 1, dose-escalation, cohorts of patients with KRAS WT advanced solid tumor malignancies will receive increasing doses of Sym015 on a Q2W schedule until establishment of the MTD or until has been evaluated. Dose-escalation will follow a standard 3+3 design with escalation dependent upon the occurrence of DLTs. The following dose levels of Sym015 will potentially be evaluated:

- Dose Level 1
- Dose Level 2:
- Dose Level 3
- Dose Level 4

An MTD may or may not be reached in the range of doses tested.

Note: Effective with protocol version 5.0 (November 2016), following review of available safety and PK data, the decision has been made to choose the following as the Q2W RP2D of Sym015: Loading dose of infused over 1.5 hours on C1/D1, followed by Q2W maintenance doses of infused over 1 hour beginning on C1/D15. As the MTD has not yet been reached, dose-escalation will continue in Part 1 of the trial to

#### Dos-Expansion Phase:

Part 2 is the Phase 2a dose-expansion portion of the study in which dosing will be at the RP2D on a biweekly (Q2W) schedule. Three cohorts will be included:

 Basket Cohort: A cohort of approximately 25 patients with KRAS WT advanced solid tumor malignancies with MET-amplification, and without available therapeutic options.
 Included in this group will be a subset of approximately 6 patients who have received prior therapy with a MET-targeting TKI.

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

CONFIDENTIAL.

Project Document Effective Date: 05Jun2019


- NSCLC MET-Amplified Cohort: A cohort of approximately 20 patients with advanced NSCLC with MET-amplification, and without available therapeutic options. Patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents.
- NSCLC MET<sup>Ex14Del</sup> Cohort: A cohort of approximately 6-12 patients with advanced NSCLC with MET<sup>Ex14Del</sup>, and without available therapeutic options. Tumors need not be MET-amplified, and patients may have received prior therapy with MET-targeting and/or EGFR-targeting agents.

During Part 2, these three cohorts will receive Sym015 at the RP2D on a Q2W dosing schedule.

The trial design is shown in Figure 1.

Overall Trial Design Part 1: Dose-escalation in KRAS WT patients Part 2: RP2D with solid framer maligrancies ading Dose followed by Standard 3+3 dose-escalation QZW Maintenauce N =12 to 15 Basket Cohort\* MET-Amplified, ERAS WT Prior MET-TKI Subset Q2W "Effective with protocol (2.0 (Dec. 2015) acround is sus **NSCLC MET-Amplified Cobort** N - 20 Q2W - --- prior MET- and/or EGFR-Targeting Agent NSCLC METERIOR Cohort Q2W N - 6 to 12 1 2 +/- MET-amplification ... prior MET- and/or EGFR-Targeting Agent Staggered enrollment between first and second patient to allow for safety assessments (Part 1) Sponsor and Investigators evaluating DLTs (Part 1), AEs and SAEs

Abbreviations: EGFR, epidermal growth factor receptor, Dec. December, KRAS, KRAS proto-oncogene; MET, MET proto-oncogene; MET exon 14 skipping alteration: N. number of patients; NSCLC, non-small cell lung carcinoma; Q2W, dosing every second week: RP2D, recommended Phase 2 dose; TKL tyrosine kinase inhibitor, WT, wild-type

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Project Document Effective Date: 05Jun2019


Symphogen A/S Sym015-01

Statistical Analysis Plan

Part 1 will be conducted in the United States (USA). Part 2 will be conducted in the USA and countries within the Asia Pacific and European regions. The number of investigational trial sites

expected to participate, will be approximately 2 to 3 in Part 1 and 15 to 27 in Part 2.

3.2 Endpoints and Associated Variables

Primary Endpoint - Part 1, Dose-Escalation

The primary objective of the dose-escalation part is to assess the safety and tolerability of Sym015.

This will be assessed by the primary endpoint for Part 1, occurrence of DLTs during Cycle 1 of

Sym015 administration.

Primary Endpoint - Part 2

The primary objective of Part 2 is to evaluate the antitumor activity of Sym015 when administered

at the Q2W RP2D. The primary endpoint is documented, confirmed OR, defined as documented

PR or CR and assessed by RECIST v1.1 at any time during trial participation by Investigator

assessment. The assessment will be performed after completion of Part 2 of the trial.

Secondary Endpoints

The following anti-tumor response endpoints will be measured in Part 1:

Documented OR, defined as documented PR or CR and assessed by RECIST v1.1 at any

time during trial participation by Investigator assessment.

Additionally, the following anti-tumor response endpoints will be measured in both Part 1 and 2:

Duration of response (DR)

Best overall response (BOR)

o SD for  $\geq$ 4 months and SD for  $\geq$ 6 months

Disease Control Rate (DCR)

o Changes in sum of diameters of target lesions from baseline to end of trial participation

 Time to disease progression (TTP) as determined based on radiological evidence

o Progression-free survival (PFS)

o Overall survival (OS)

### 3.2.1 Efficacy Variables

3.2.1.1 Tumor evaluation and time to event variables

The anti-tumor activity of Sym015 will be assessed by the Investigator, or qualified designee, according to RECIST v1.1 [6].

Patients will undergo imaging by CT or MRI of neck, chest, abdomen and pelvis as indicated based on tumor type and clinical judgment in order to follow the underlying malignancy. The use of CT or MRI must be consistent per patient throughout the trial.

Screening

Note: A CT/MRI performed within 28 days prior to Day 1 may be used for evaluation of eligibility and as baseline scan, provided that the CT/MRI has been performed according to the protocol requirements

• EOC2 and end of every second cycle thereafter, i.e., EOC4, EOC6, EOC8, etc.

Note: May be performed at any time during the week prior to Day 1 of the next cycle, including Day 1 of the next cycle, prior to dosing (provided results are available prior to study drug administration)

Suspected PD (as soon as possible)

• At least 28 days following an OR (PR, CR)

EOT (if >3 weeks since previous CT/MRI)

At 1M FUP (if PD was not documented before or at EOT)

If PD is documented at any time, no further disease assessments will be required. Patients with documented PD will be discontinued from Sym015 so that alternative management of their malignancy may be considered.

For all imaging time points, the following will be recorded as per RECIST v1.1: Target lesions including size, location, and type (nodal/non-nodal); sum of diameters of target lesions; any new lesions noted during trial, including size, location, and type (nodal/non-nodal); final response assessment at each visit (PD, SD, PR, CR or Not Evaluable [NE]), per investigators evaluation.

Tumor evaluation according to RECIST 1.1 will be the basis for the derivation of all efficacy endpoints.

To be assigned a status of PR or CR, changes in disease status must be confirmed by repeat imaging studies performed no less than 28 days (4 weeks) after the criteria for response are first met. In the case of SD, follow-up measurements must have met the SD criteria at least once after trial entry at a minimal interval in general no less than 6-8 weeks from first dose of Sym015; for the scope of derivation of SD as BOR, a minimal SD duration of 6 week will be required.

The following anti-tumor response endpoints will be derived based on Tumor evaluation according to RECIST 1.1:

Target and Non-target Response at each timepoint will be derived according to RECIST 1.1 [6].

> o Evaluation of target lesions will be derived based on sum of diameters as follow:

'Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

TP-GDO-WW-133-01

Effective Date: 05 Sep 18

Related to: SOP-GDO-WW-019


Symphogen A/S Sym015-01

Statistical Analysis Plan

 Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or

more new lesions is also considered progression).

 Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest

sum of diameters while on study.'

 Evaluation of non-target lesions: non-target lesions response will be reported in CRF as CR, NON-CR/NON-PD, PD, Not Evaluated; worst response will be taken as the Non-Target Lesion response for the correspondent timepoint; for assessment of worst response the following order will be followed: PD, Not

Evaluated, NON-CR/NON-PD, CR.

Target and Non-Target Response at each timepoint, derived as described, will be reviewed

by Symphogen and a patient by patient basis across time.

At each timepoint Overall Responses will be captured in CRF; as well Overall Responses will also be derived according to RECIST 1.1 [6]: Table 1 of above-mentioned paper [6] reported below is reflected in CSP Table 14 'Overall Response Status for Patients with Baseline Measurable Disease' and will be used to derive overall response at each time point for patients who have measurable disease at baseline. When patients have non-measurable (therefore non-target) disease only, Table 2 is to be used.

Overall responses derived as described are supposed to coincide with overall responses collected in CRF; cases of mismatch will be queried; any unsolved case of mismatch will be reviewed by Symphogen and the suppose of mismatch by patient basis across time.

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 CONFIDENTIAL

Table 1 - Time point response: patients with target (+/non-target) disease.

| Target lesions | Non-target lesions | New<br>lesions | Overall<br>response |
|---|---|---|---|
| CR | CR | No | |
| CR | Non-CR/non-PD | | CR |
| CR | Not evaluated | No | PR |
| PR | | No | PR |
| • | Non-FD or | No | PR |
| SD | not all evaluated<br>Non-PD or<br>not all evaluated | No | SD |
| Not all<br>evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| łπy | PD | Yes or No | |
| Any | Any | Yes | 6D<br>6D |

CR = complete response, PR = partial response, SD = stable disease.

Eisenhauer EA, Therasse P, Bogaerts J, et al: New response evaluation criteria in solid tumors: Revised RECIST guideline

Table 2 - Time point response: patients with non-target

| Non-target lesions | New lesions | Overall response |
|---|---|---|
| CR<br>Non-CR/non-PD<br>Not all evaluated<br>Unequivocal PD<br>Any | No<br>No<br>No<br>Yes ar No | CR<br>Non-CR/non-PD <sup>2</sup><br>NE<br>PD |
| CR = complete response,<br>NE = inevaluable. | Yes<br>PD = progressive | PD<br>disease, and |

a 'Non-CR/non-PD' is preferred over 'stable disease' for non-target disease since SD is increasingly used as endpoint for assessment of efficacy in some trials so to assign this category when no

Eisenhauer EA, Therasse P, Bogaerts J, et al: New response evaluation criteria in solid tumors: Revised RECIST guideline (version 1.1). Eur J Cancer 2009; 45:228-247

# Best overall response (BOR)

The best overall response is determined once all the data for the patient is known. Patients with non-target disease only, may have a time point response of NON-CR/NON-PD, these responses will be considered as SD for derivation of BOR.

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

CONFIDENTIAL Project Document Version No. 1.0 Project Document Effective Date: 05Jun2019


PD = progressive disease, and NE = inevaluable.

lesions can be measured is not advised.

Determinations of BORs derived as here described will be reviewed by Symphogen and on a patient by patient basis across time.

The best overall response is the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation. Specifically, in non-randomised trials where response is the primary endpoint, confirmation of PR or CR is needed to deem either one the 'best overall response'. [6]

When a CR or PR is achieved but is not confirmed at subsequent assessment time point, the BOR will be reported as unconfirmed CR or PR.

Best response determination in trials where confirmation of complete or partial response is required: Complete or partial responses may be claimed only if the criteria for each are met at a subsequent time point as specified in the protocol. [6]

Employed rules for CR/PR BOR derivation are schematically reported in below Table 3.

| Table 3 – Rules for Complete and Partial Response BOR derivation | | |
|---|---|---|
| Overall response at timepoint | Overall response<br>Subsequent<br>timepoint | BOR |
| CR | CR | Confirmed CR |
| CR | PR | Unconfirmed CR |
| CR | SD | Unconfirmed CR |
| CR | PD | Unconfirmed CR |
| CR | NE | Unconfirmed CR |
| PR | CR | If subsequent overall response is CR: Confirmed CR If subsequent overall response is not CR: Confirmed PR |
| PR | PR | Confirmed PR |
| PR | SD | Unconfirmed PR |
| PR | PD | Unconfirmed PR |
| PR | NE | Unconfirmed PR |

Symphogen A/S Sym015-01

Statistical Analysis Plan

Should a patient have responses of unconfirmed CR and confirmed PR, BOR will be defined as confirmed PR for that patient.

When SD is believed to be best response, it must also meet the protocol specified minimum

time from baseline (specified as 6 weeks in this trial). If the minimum time is not met when

SD is otherwise the best time point response, the patient's best response depends on the

subsequent assessments. For example, a patient who has SD at first assessment, PD at

second and does not meet minimum duration for SD, will have a best response of PD. The

same patient lost to follow-up after the first SD assessment would be considered NE.

Documented Objective Response (OR), is defined as confirmed CR or PR, based on

determination of confirmed BOR.

Duration of response (DR)

The duration of overall response is measured from the time measurement criteria are first

met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive

disease is objectively documented (taking as reference for progressive disease the smallest

measurements recorded on study). '[6].

Duration of Response (weeks) = (Date of PD or Death [whichever is first recorded] - Date

of first CR/PR [whichever is first recorded] + 1) / 7

Duration of Response will be presented at one decimal place precision.

In case of patients out of study before experiencing PD or death, the duration of response

will be measured up to the last available valid tumor assessment per RECIST v1.1.

Changes in sum of diameters of target lesions from baseline For patients with measurable

disease (i.e., with target lesions), absolute and percent changes in the sum of diameters of

target lesions from baseline will be calculated, the best change will be identified as the

nadir, i.e. largest reduction or smallest increase. This endpoint will not be derived for

patients who do not have a baseline tumor assessment or who do not have any post-baseline

tumor assessments.

Time to disease progression (TTP) as determined based on radiological evidence

Time to documented PD (based on radiological assessments) will be derived and expressed in the unit of weeks. TTP is defined as the time from first dose of study drug until objective tumor progression; TTP does not include deaths [7]. Based on this definition, PD will be counted as outcome; patients with last tumor assessment showing CR or PR or SD will be censored at the time of last available tumor assessment per RECIST v1.1; patients who died for any causes (including deaths of disease but with no documented PD) will be censored at the time of last available tumor assessment per RECIST v1.1.

TTP (weeks) = (Date of PD – Date of first IMP infusion + 1)  $\frac{7}{7}$ 

SD for  $\geq$  months and SD for  $\geq$ 6 months

'Stable disease is measured from the start of the treatment (in randomised trials, from date of randomisation) until the criteria for progression are met, taking as reference the smallest sum on study (if the baseline sum is the smallest, this is the reference for calculation of PD). '[6].

Therefore, determination of SD duration ≥4 months and ≥6 months will be based on the calculated value of TTP regardless of censoring. If a month corresponds to 4.34524 weeks, a TTP of 17.381 will be needed to claim an SD duration ≥4 months; as well, a TTP of 26.0715 will be needed to claim an SD duration ≥6 months

Disease control rate (DCR)

The DCR is defined as the percentage of patients who had BOR of confirmed CR or confirmed PR or SD (including unconfirmed CR/PR, provided 6 weeks minimum criteria for SD duration is met).

Progression Free Survival (PFS)

PFS is defined as the time from first dose of study drug until objective tumor progression as determined based on radiological evidence or death, whichever occurs first [7]. PFS data

will be censored on the date of the last adequate tumor assessment for patients who do not TP-GDO-WW-133-01

have an event (PD or death) at data cutoff, or for patients who died after two or more subsequent missing response assessments (which correspond to 63 days considering 2 times the 28-days scheduled time interval between two subsequent response assessments, plus 7 days' time window). Patients who do not have a baseline tumor assessment or who do not have any post-baseline tumor assessments will be censored at start of treatment unless death occurred, in which case the death will be considered an event.

PFS (months) = (Date of PD or Death [whichever is first recorded] - Date of first IMP infusion + 1) / 30.4375.

Moreover, for the scope of an additional sensitivity analysis, non-radiological clinical progression will also be considered as an outcome; date of clinical progression is available in CRF at end of treatment page.

Overall Survival (OS)

Overall survival is defined as the time from first dose of study drug until death from any cause. After the 1M FUP Visit, the Investigator will make every effort to obtain follow-up information on response assessment and/or overall survival (OS) about once every 2 months. Survival follow-up is required until death, withdrawal of consent, trial site closure, or termination/end of the trial. Occurrence of one of these events constitutes the EOS for the patient. Patients alive at EOS will be censored at the time of last contact when patient is known to be alive.

OS (months) = (Date of Death – Date of first IMP infusion + 1) / 30.4375

3.2.1.2 Pharmacodynamic Variables

These variables include:

Tumor Markers Evaluation (Part 1 and Part 2 Basket Cohort) recommended to be evaluated at timepoints coinciding with the CT/MRI

Archival Tumor Tissue for MET and KRAS assessment (Part 1 and Part 2 Basket Cohort)

collected at Screening; if archival tissue is not available, tissue from a tumor biopsy TP-GDO-WW-133-01 CONFIDENTIAL

Symphogen A/S Sym015-01

Statistical Analysis Plan

performed during screening is used; assessment of MET-amplification status is optional in

Part1.

Tumor Biopsy for Eligibility Assessment (Part 1 and Part 2 Basket Cohort) collected at

Screening

Tumor Biopsy for Biomarkers Analysis

o Part 1: only applicable for patients with known MET-amplification who consent to this

optional procedure. Collected at Screening, at End of Cycle (EOC) 2 (i.e., coinciding

with time of first response assessment) or upon PD, whichever occurs first

o Part 2 Basket Cohort: Required at Screening if archival tissue is unavailable or

insufficient for central analysis (to be performed after confirmation of eligibility);

Required at End of Cycle 2 (i.e., coinciding with time of first response assessment) or

upon PD, whichever occurs first

o Part 2 NSCLC<sup>Ex14Del</sup> Cohort: optional at Screening and at EOC 2 (i.e., coinciding with

time of first response assessment) or upon PD, whichever occurs first

o Part 2 NSCLC MET-Amplified Cohort: required at Screening; Optional at EOC 2 (i.e.,

coinciding with time of first response assessment) or upon PD, whichever occurs first

Tumor Biopsy for MET Status

o Part 2 NSCLC MET-Amplified Cohort: Required at Screening, tissue from a newly

performed pre-dosing tumor biopsy must be submitted for central confirmation of

MET-amplification; Optional at EOC 2 (i.e., coinciding with time of first response

assessment) or upon PD, whichever occurs first

o Part 2 NSCLC<sup>Ex14Del</sup> Cohort: Required at Screening, tissue from a recent or newly

performed pre-dosing tumor biopsy must be submitted for central assessment of

METEx14Del; Optional at EOC 2 (i.e., coinciding with time of first response

assessment) or upon PD, whichever occurs first

Related to: SOP-GDO-WW-019


Symphogen A/S Sym015-01

Statistical Analysis Plan

• Blood Sample for Genomic and Biomarker Analyses: Screening (it will be permissible to

perform this procedure outside the 14-day screening period, provided informed consent for

the trial has been obtained); EOC 2 (coinciding with time of first response assessment or

upon PD, whichever occurs first); End of Treatment (if after EOC 2; need not repeat if

patient is discontinuing at the EOC 2 or if a sample was obtained upon PD)

• Skin biopsy (Part 1 only): Screening, EOC2 (i.e., coinciding with time of first response

assessment) or upon PD, whichever occurs first

3.2.1.3 Immunogenicity Variables

Anti-drug antibody (ADA) Testing: all samples must be taken prior to the Sym015 infusion of that

visit. Analysis of ADA and residual serum levels of Sym015 will be performed at a specialty

laboratory. ADA samples are collected are C1/D1, C2/D1 (Part 2 only), Day 1 of every second

cycle thereafter, i.e., Cycle 3, 5, 7 etc. (prior to dosing), EOT, 1M FUP.

3.2.2 Pharmacokinetic Variables

Derivation of PK parameters will be the responsibility of Symphogen A/S.

PK samples will be taken according to the schedules shown in CSP Table 9. The serum

concentration of Sym015 is defined as the sum of the serum concentration of the two constituent

antibodies of Sym015, Hu9006 and Hu9038-

The PK endpoints will be derived based on the serum concentration versus time curves of Sym015,

and the first infusion of Sym015 in both parts of the trial. Refer to CSP Table 11.

C<sub>max</sub>, C<sub>trough</sub> and T<sub>max</sub> will be derived from observed data while AUC<sub>1</sub>, AUC<sub>norm, 7</sub>, CL, V<sub>z</sub>, and T<sub>1/2</sub>

will be estimated using non-compartmental methods and actual time points.

Table 9 Schedule of Pharmacokinetic Assessments

| | Window | Cycle 1 | | | Cycles Thereafter | | EOT | IM FUP |
|---|---|---|---|---|---|---|---|---|
| Sampling Time | | D1-D3 | D8 | D15 | Dl | D15 | | |
| Part 1 / Part 2 B | asket Cohor | | 7 | | | | | |
| Prior to SOI | -4h | X | | $X^{1}$ | X3 | $X^1$ | | |
| EOI | - 10 min | X | | X2 | $X^{i}$ | $X^{2}$ | | |
| EOI + 1 h | ±15 min | X | | | | | | |
| EOI + 2 h | ±30 min | X | | | | | | |
| EOI ÷ 4 h | ±30 min | X | | | | | | |
| EOI÷Sh | ±90 min | X | | | | | | |
| EOI + 24 h | ≐ố h | X | | | | | | |
| EOI ÷ 48 h | =12 h | X | | | | | | |
| During Visit | NA | | X | | | | X | X |
| Part 2 NSCLC ( | oborts (effe | ctive with p | rotocol | 3.0; Dec | ember 2018 | ) | | |
| Prior to SOI | -4h | X | | X: | $X_3$ | $X^1$ | | |
| EOI | - 10 min | X | | $X^{i}$ | $X^2$ | X: | | |
| EOI+4h | ±30 mm | X | | | | | | |
| EOI ÷ 48 h | =12 h | Х | | | | | | |
| During Visit | NA | | X | | | | X | X |

Abbreviations (in high-benned order), D. day, EOI, End of Infusion. EOT, End of Treatment Visit, NA, Not Applicable, E. hour, minutes, IM FUP, 1-Month Follow-up Visit, SOI, Start of Infusion.

1) ESymo15 is possed, only one PEI sample should be taken during the visit.

Table 11 PK Endpoints Definitions and Derivations

| Symbol | Definition and derivation |
|---|---|
| Cxongh | Trough concentration (i.e., concentration of Sym015 measured pre-infusion) |
| AUC, | Area under the concentration-time curve in a dosing interval (i.e., from time zero (end of infusion) up to 336 hours or 504 hours depending on regimes). AUC, will be calculated using the linear trapezoidal method and interpolated in case of measurements after 336/504 hours, or extrapolated using terminal rate constant and the last quantifiable concentration. C <sub>2</sub> |
| C <sub>2</sub> | Last quantifiable concentration. C <sub>x</sub> is not an endpoint, but is used for derivation of endpoints |
| AUC | Dose normalized area under the concentration-time curve in a dosing interval, calculated as AUC; divided by the dose infused |
| C | Maximum concentration |
| Tana | Time to reach maximum concentration |
| Ã.z | Terminal rate constant (negative of the slope of an Inlinear regression of the un-weighted data considering the terminal phase of the concentration-lime curve $\geq$ limit of quantification. $\lambda_z$ is not an endpoint, but is used for derivation of endpoints |
| Γ-, | Terminal elimination half-life, calculated as ln(2); \(\lambda_a\) |
| CL | Clearance (Dose/AUC.) |
| $V_z$ | Volume of distribution during the terminal phase $(CL/\lambda_z)$ |

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

Project Document Effective Date: 05Jun2019


### 3.2.3 Safety Variables

- Medication/Procedure Survey
- Adverse Events (AE) Survey
- Dose-Limiting Toxicities Evaluation (Part 1 Only)
- Vital Signs and Body Weight
- Performance Status
- Physical Examinations
- Electrocardiograms (ECG)
- Echocardiogram (ECHO) or Multi-Gated Acquisition Scan (MUGA)
- Clinical Laboratory Assessments and Pregnancy Test

### 3.2.3.1 Medication/Procedure Survey

To include all medications taken other than Sym015 and all procedures performed during trial. For medications the following are collected: generic name or brand name, indication for use, dose and frequency, route of administration, start and stop dates or if ongoing at 1M FUP Visit. For procedures the following are collected: date and reason for procedure.

Collected starting from the date of Screening and until the date of the 1M FUP.

Full description and analysis are detailed in section 4.8.

### 3.2.3.2 Adverse Events (AE) Survey

All AEs will be recorded from signing of informed consent for participation in the trial. The recording period ends at the time of the 1M FUP Visit. All AEs should be followed until they are resolved or until the 1M FUP Visit, whichever comes first.

Definition of AE

Symphogen A/S Sym015-01

Statistical Analysis Plan

An AE is any untoward medical occurrence in a patient or a clinical investigation Patient

administered a pharmaceutical product, and which does not necessarily have a causal relationship

with this treatment. An AE can therefore be any unfavorable and unintended sign (including an

abnormal laboratory finding), symptom, or disease temporally associated with the use of an IMP,

whether or not considered related to the IMP.

Causality for the above-mentioned AE will be assessed appropriately by the investigator as

detailed below in this paragraph.

A pre-existing condition (i.e., a disorder that is present before the AE recording period starts and

is noted on the medical history/physical examination form) should not be recorded as an AE unless

the condition worsens, or episodes increase in frequency during the AE recording period.

PD will not be captured as an AE unless the nature of the PD is different than expected (i.e., other

diagnosis and/or signs/symptoms that are not typical of PD) as assessed by the Investigator.

Definition of Treatment-emergent AE (TEAE)

Treatment-emergent AEs (TEAEs) are events that occur on or after first dose of the study

medication or a worsening in severity of a pre-existing condition occurring after first dose of the

study medication.

Definition of Infusion Related Reaction (IRR)

An IRR is defined as an AE occurring during the Sym015 infusion and up to 2 hours after the end

of infusion (EOI), which is assessed by the Investigator to be related to the infusion of Sym015.

Signs of IRRs may include but are not limited to facial flushing and swelling, shortness of breath,

headache, diaphoresis, tachycardia, hypotension, chills, rigors, chest and throat tightness, as well

as chest, back and/or abdominal discomfort. If an IRR occurs, it should be classified according to

the Common Terminology Criteria for Adverse Events (Version 4.03) (CTCAE v4.03). In all

cases, the Investigator should use best clinical judgment in managing such reactions.

All IRRs must be reported in the CRF as an AE with the term "Infusion-related Reaction" followed

by a specification of symptoms (e.g., "Infusion-related Reaction with dyspnea and flushing").

Symphogen A/S Sym015-01

Statistical Analysis Plan

Definition of AE duration

AE duration will be derived as AE duration = (AE end date - AE onset date +1); in case of AE

ongoing, the date of last contact with the patient will be used as AE for the scope of derive the AE

duration.

Definition of Serious AE (SAE)

An SAE is an AE that meets one or more of the following outcome criteria:

Results in death

Is life-threatening (patient is at immediate risk of death at the time of the event; it does not

refer to an event which hypothetically might cause death if it was more severe)

Requires inpatient hospitalization or prolongation of existing hospitalization

Results in persistent or significant disability/incapacity

Is a congenital anomaly/birth defect

• Is medically important (Medically important events may not be immediately life-

threatening or result in death or hospitalization but may jeopardize the patient or may

require intervention to prevent one of the other outcomes listed in the definition above).

AE Severity

The Investigator will use the CTCAE v4.03 to describe the severity of an AE. If the severity of an

AE is not specifically graded by the CTCAE guidance document, the Investigator should use the

general definitions of Grades 1 to 5 as per the following, and use his/her best medical judgment to

describe the severity of the AE:

Grade 1: Mild

Grade 2: Moderate

Grade 3: Severe

Symphogen A/S Sym015-01

Statistical Analysis Plan

Grade 4: Life-threatening or disabling

Grade 5: Death caused by the event

Changes in severity of AEs will be recorded.

AE Relationship to IMP

The Investigator must assess causal relationship to the IMP, Sym015. The causal relationship is an assessment of whether or not the event is related to the use of the IMP. It is not an evaluation of whether or not the event could hypothetically occur in the investigational patient population.

The causal relationship of an AE to the IMP, Sym015, will be rated as follows:

Not Related: The AE is not related to the IMP, which means the event:

o Does not follow a reasonable temporal sequence from drug administration

o Is readily explained by the patient's clinical state or by other modes of therapy

administered to the patient

The AE is clearly NOT related to the IMP

• Unlikely Related: The AE is considered not related to the IMP based on the following:

o Does not follow a reasonable temporal sequence from administration of drug

o Could readily be a result of the patient's clinical state, environmental, or toxic factors,

or other modes of therapy

Does not follow a known response pattern to the suspected drug

Does not reappear or worsen when the drug is re-administered

Possibly Related: The AE might not be related, but possibility cannot be ruled out with

certainty and therefore would be considered related based on:

Follows a reasonable temporal sequence from administration of drug

- Could readily have been a result of the patient's clinical state, environmental or toxic factors, or other modes of therapy
- o Follows a known response pattern to the suspected drug
- Probably Related: It has been determined with a high degree of certainty that the AE is associated with administration of IMP based on:
  - o Follows a reasonable, temporal sequence
  - Cannot be reasonably explained by known characteristics of the patient's clinical state, environmental, or toxic factors, or other modes of administered therapy
  - The AE disappears or decreases in severity upon cessation of drug, or reduction in dose.
  - Follows a known response pattern to the suspected drug
- Related: The AE is related to the IMP, which means the event:
  - o Follows a reasonable temporal sequence from drug administration
  - o Abates upon discontinuation of the IMP (de-challenge)
  - Is confirmed by reappearance of the reaction on repeat exposure (re-challenge)
  - Cannot be reasonably explained by the known characteristics of the patient's clinical state
  - Is not likely to have been produced by the patient's clinical state or by other modes of therapy administered to the patient

## **Outcome**

Outcome of the AE must be assessed by the Investigator utilizing one of the following terms:

- Recovered
- Recovered with sequelae (if recovered with sequelae, specify sequelae)

Symphogen A/S Sym015-01

Statistical Analysis Plan

Not recovered

Fatal

Unknown

Instructions for reporting changes in an ongoing AE during a patient's participation in the trial are provided in the instructions that accompany the AE CRF pages.

Handling of partial AE onset and end date

Any AEs with incomplete start and end dates will be treated as follows:

• Adverse events with completely unknown onset date will be considered as treatment-

emergent; for the scope of AE duration derivation, these AE will be considered as occurred

the day of first IMP infusion.

Adverse events with unknown start day and month but with known start year will be

considered:

o as treatment-emergent if the start year coincides or is after the first dosing year; for the

scope of AE duration derivation, these AE will be considered as occurred the day of

first IMP infusion if the start year coincides with first dosing year, as occurred on 1st

January otherwise (i.e. in case the start year is after the first dosing year)

o as non-treatment emergent if start year is before the first dosing year; for the scope of

AE duration derivation, these AE will be considered as occurred on 1<sup>st</sup> January.

Adverse events with unknown start day but with known start month and year will be

considered:

o as treatment-emergent if the start month and year coincide or are after the month and

year of first dosing; for the scope of AE duration derivation, these AE will be

considered as occurred the day of first IMP infusion if the start month and year

coincides with first dosing month and year, as occurred on 1st day of the month

otherwise (i.e. in case the month and year is after the month and year of first dosing)
Symphogen A/S Sym015-01

Statistical Analysis Plan

o as non-treatment emergent if start month and year is before the month and year of first dosing; for the scope of AE duration derivation, these AE will be considered as

occurred on 1st day of the month.

Adverse events with completely unknown end date will be considered as ended on the day

of last contact with the patient).

Adverse events with unknown end day and month but with known end year:

o if the AE end year if before the year of last contact with the patient, AE will be

considered as ended on 31th December.

o if the AE end year coincide with the year of last contact with the patient, AE will be

considered as ended on day of last contact with the patient.

o If AE end year is after the year of last contact with the patient, for the scope of derive

the AE duration the date of last contact with the patient will be used as AE end date.

Adverse events with unknown end day but known end month and end year:

o if the AE end month and year are before the month and year of last contact with the

patient, AE will be considered as ended on last day of the month.

o if the AE end month and year are coinciding with the month and year of last contact

with the patient, AE will be considered as ended on last day of last contact with the

patient.

o If AE end month and year are after the month and year of last contact with the patient,

for the scope of derive the AE duration the date of last contact with the patient as AE

end date.

Adverse events with completely or partial unknown start and end dates will be shown as not known


(NK), for the respective unknown part, in the listings.

3.2.3.3 Dose-Limiting Toxicities Evaluation (Part 1 Only)

A DLT is defined as any of the following toxicities that occur during the DLT observation period, if considered related (causality rating of possibly, probably, or related) to Sym015:

- 1. Grade 3 non-hematologic toxicity regardless of duration, with the exceptions of:
  - a. Grade 3 nausea, vomiting, diarrhea, or fatigue lasting  $\leq$  2 days with best supportive care
  - b. Grade 3 asymptomatic electrolyte abnormalities lasting  $\leq$  3 days that are not considered clinically relevant by the Investigator and that resolve with medical therapy
- 2. Any Grade 4 non-hematologic toxicity, with the exception of:
  - a. Grade 4 asymptomatic electrolyte abnormalities lasting < 3 days that are not considered clinically relevant by the Investigator and that resolve with medical therapy.
- 3. Neutropenia that is:
  - a. Grade 3-4 febrile neutropenia
  - b. Grade 4 and sustained (i.e., ANC <500 per mm3, duration >5 days)
- 4. Thrombocytopenia that is:
  - a. Grade 3 with clinically significant hemorrhage
  - b. Grade 4 (platelets < 25,000 per mm3)
- 5. AST/ALT elevation > 3xULN with bilirubin elevation > 2xULN that cannot be explained by factors not related to study drug
- 6. Inability to complete Cycle 1 at the assigned dose due to  $\geq$  Grade 3 toxicity
- 7. Treatment delays >2 weeks from the scheduled "next dose" due to  $\ge$  Grade 3 toxicity

DLT events (Yes / No) are collected in CRF as well as date of assessment, DLT description and AE Reference.

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 CONFIDENTIAL

Project Document Effective Date: 05Jun2019


Symphogen A/S Sym015-01

Statistical Analysis Plan

The observation period for DLTs is defined as Cycle 1 with a final assessment 14 (±2) days after

the last dose of Cycle 1 or prior to dosing on C2/D1.

Cycle 1 must have been completed at the assigned dose of Sym015 for a patient to complete the

DLT observation period.

3.2.3.4 Vital Signs and Body Weight

To include temperature, heart rate, blood pressure, and body weight. Collected at Screening, Prior

to each dosing, at EOT, at 1M FUP and as clinically indicated

3.2.3.5 Performance Status

To be assessed by Eastern Cooperative Oncology Group (ECOG) performance Status (PS) score.

Collected at Screening, at Day 1 of each cycle (prior to dosing; does not need to be assessed prior

to C1/D1 if assessed during screening  $\leq 7$  days from C1/D1), at EOT, at 1M FUP and as clinically

indicated.

**ECOG PS Score:** 

0=Fully active, able to carry on all pre-disease activities without restrictions

• 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of

a light or sedentary nature e.g., light housework, office work

2=Ambulatory and capable of self-care, but unable to carry out any work activities. Up

and about more than 50% of waking hours

• 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking

hours

4=Completely disabled. Cannot carry on self-care. Totally confined to bed or chair

5=Dead

Symphogen A/S Sym015-01

Statistical Analysis Plan

3.2.3.6 Physical Examination

To include evaluation of the following at Screening: General appearance, skin, head, ears, eyes,

nose, throat, neck/thyroid, chest, cardiovascular system, abdomen, musculoskeletal system, lymph

nodes, neurologic status, and mental status; include height (without shoes, rounded to nearest

centimeter). Thereafter, a targeted physical examination may be performed as indicated.

To be assessed at Screening, at Day 1 of each cycle (prior to dosing; does not need to be performed

prior to C1/D1 if performed during screening ≤ 7 days from C1/D1), at EOT, at 1M FUP, and as

clinically indicated.

3.2.3.7 Electrocardiograms (ECG)

A 12-lead ECG will be performed on Screening, EOT, and as clinically indicated.

Parameters measured will include heart rate, PR, R-R, QRS, QT, and QTc intervals (calculated by

the Fridericia [QTcF] or Bazzett's [QTcB] correction formula). Clinical assessment (abnormality

as clinically significant or not clinically significant) will be performed.

3.2.3.8 Echocardiogram (ECHO) or Multi-Gated Acquisition Scan (MUGA)

ECHO or MUGA scan will be performed at Screening, in the event of cardiac symptoms (e.g.,

shortness of breath, edema) and as otherwise clinically indicated.

3.2.3.9 Clinical Laboratory Assessments and Pregnancy Test

Blood samples will be taken at all scheduled visits and will be analyzed for the following

parameters as per CSP Table 8 and as clinically indicated:

Table 8 Schedule of Safety Blood and Urine Samples

| Sample Analysis Day within Cycle | Screening | Cycle 1 | | | | Cycles<br>Thereafter | | EOT | IM<br>FUP |
|---|---|---|---|---|---|---|---|---|---|
| | | DI | D3<br>D8 | D15 | D22 | D1 | D15 | | |
| Hematology Panel | X | $-X_{\rm L}$ | X | Х | Х | X | Х | Х | 3. |
| Biochemistry Panel | X | $-\Sigma_1$ | X | X | X | X | X | X | X |
| Coagulation Panel | X- | $X_1$ | : 1 | X | X | X | X | X | X |
| Urmalysis | Z | $-X^{t}$ | | X | | X | | X | X |
| Pregnancy Test | Z | | | | | | | X | i |

Abbreviations (in alphabetical order); D. day, EOT, End of Treatment Visit IM FUP, I-Month Follow-up Visit

- Hematology panel (complete blood count with differential, ANC, and platelet count): at Screening, Cycle 1 (weekly prior to dosing if on dosing day, Day 3. Note: Does not need to be performed prior to C1/D1, if performed during screening ≤7 days from C1/D1), each cycle thereafter (Day 1 and 15 prior to dosing), EOT, 1M FUP, and as clinically indicated.
- Biochemistry panel (sodium, potassium, chloride, bicarbonate or carbon dioxide, blood urea nitrogen (BUN), creatinine, glucose, bilirubin [total and direct], AST, ALT, ALP, calcium, magnesium, phosphorus, albumin, total protein, uric acid, amylase, lipase, and creatine kinase): at Screening, Cycle 1 (weekly prior to dosing if on dosing days, Day 3. Note: Does not need to be performed prior to C1/D1, if performed during screening ≤7 days from C1/D1), each cycle thereafter (Day 1 and 15 prior to dosing), EOT, 1M FUP, and as clinically indicated.
- Coagulation panel (PT, PTT and INR): at Screening, Cycle 1 (Day 1 and 15 prior to dosing.
  Note: Does not need to be performed prior to C1/D1, if performed during screening ≤7
  days from C1/D1), each cycle thereafter (Day 1 prior to dosing), EOT, 1M FUP, and as clinically indicated.
- Urinalysis (specific gravity, pH, protein, glucose, ketones, occult blood, leukocyte esterase, nitrite, bilirubin, and urobilinogen): at Screening, Cycle 1 (Day 1 and 15 prior to dosing. Note: Does not need to be performed prior to C1/D1, if performed during screening ≤7 days from C1/D1), each cycle thereafter (Day 1 prior to dosing), EOT, 1M FUP, and as clinically indicated.

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


<sup>1)</sup> Does not need to be performed prior to C1 D1 if performed during screening 27 days from C1/D3

Symphogen A/S Sym015-01

Statistical Analysis Plan

• Pregnancy test (serum human Chorionic Gonadotropin (β-hCG) at screening, urine β-hCG

thereafter, in women of childbearing potential): at Screening, EOT and as clinically

indicated.

All clinical laboratory test results will be graded per NCI CTCAE v4.03 if applicable, as well as

high (higher than the normal range), normal (in the normal range) and low (lower than normal

range).

4 STATISTICAL METHODS

4.1 Data Quality Assurance

All tables, figures and data listings to be included in the report will be independently checked for

consistency, integrity and in accordance with standard procedures.

4.2 General Presentation Considerations

4.2.1 Baseline

'Baseline' is defined as the last available pre-treatment assessment, considering both scheduled

and unscheduled assessments.

Safety assessments at Cycle 1 Day 1 with no time of assessment (i.e. Vital Signs and Body Weight,

ECOG PS, Physical Examination) are assumed to be taken pre-treatment.

4.2.2 End of Treatment (EOT)

'End of Treatment' is defined as the first assessment obtained on or after the last dose of study

treatment, considering both scheduled and unscheduled assessments.

4.2.3 Unscheduled assessments

Unscheduled assessments will be presented in listings in chronological order.

By-visit summaries of each test/exam will be tabulated according to the protocol defined visit

schedule.


Post Baseline safety unscheduled assessments (for Clinical Laboratory, ECG QTc, etc.) will be used for determination of worst result (i.e. Maximum and Minimum post Baseline result) as well as the maximal laboratory CTCAE grade if applicable; also, all post baseline tumor evaluation assessments will be used to derive BOR.

Moreover, post baseline, worst by-visit result will be used in by-visit summaries of Clinical Laboratory. In this case, both scheduled and unscheduled results will be used to determinate worst by-visit result. Each unscheduled result will be bracketed into scheduled visits. Sites should define which scheduled timepoint each unscheduled laboratory assessments belongs to; this information is captured in CRF. In the case such information will not be available, following rules will apply:

- safety blood laboratories obtained after first dosing and up to C1D5 will be bracketed in C1D3;
- o safety blood laboratories obtained from C1D6 up to C1D10 will be bracketed in C1D8;
- safety blood laboratories obtained from C1D11 up to pre-dose on the day of Cycle 1 second infusion will be bracketed in C1D15;
- safety blood laboratories obtained from post-dose on the day of Cycle 1 second infusion up C1D24 will be bracketed in C1D22
- o safety blood laboratories obtained from C1D25 to pre-dose on the day of Cycle 2 first infusion will be bracketed in C2D1;
- o safety blood laboratories obtained from post-dose on the day of Cycle 2 first infusion up to pre-dose on the day of Cycle 2 second infusion will be bracketed in C2D15;
- o safety blood laboratories obtained from post-dose on the day of Cycle 2 second infusion up to pre-dose on the day of Cycle 3 first infusion will be bracketed in C3D1;
- Starting from C3, safety blood laboratories obtained from post-dose on the day of the previous Cycle second infusion up to pre-dose on the day of the current Cycle first infusion will be bracketed in the current Cycle D1;

Related to: SOP-GDO-WW-019

 Starting from C3, safety blood laboratories obtained from post-dose on the day of the current Cycle first infusion up to pre-dose on the day of current Cycle second infusion will be bracketed in the current Cycle D15;

Safety blood laboratory result associated with higher CTCAE grade by visit, will be flagged as worst by visit result and used in by visit summary tables; if multiple within visit unscheduled results are associated with the same CTCAE grade, the most extreme value in the direction used for CTCAE grade derivation will be flagged as the worst. Safety blood laboratory test for which a CTCAE grade derivation rule is not available, the by visit result farthest to the normal range limit will be flagged as worst by visit result and used in by visit summary tables; results above normal ranges will be compared with upper limit of normality, while results below normal ranges will be compared with lower limit of normality; it is not expected to observe in the same visit abnormal high and low results, should this occur the worst within visit will be manually flagged after data review from medical perspective. In case all by visit results are within normal ranges and not associated with a CTCAE grade, or in case no CTCAE and no normal ranges are available for a specific parameter, result obtained at the scheduled assessment will be used in the by visit summary tables and if no scheduled assessment is available the by visit unscheduled closest to the scheduled timepoint will be considered.

Except considered as Baseline, EOT or worst result or worst by visit result for safety blood laboratories, unscheduled assessments will not be included in summaries.

#### 4.2.4 Treatment Day

'Treatment Day' will be calculated relative to the date of C1/D1 as follow:

assessments taken before the first infusion of IMP

Treatment Day = Assessment Date - First IMP infusion Date

assessments after the first infusion of IMP

Treatment Day = Assessment Date - First IMP infusion Date + 1.

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

Symphogen A/S Sym015-01

Statistical Analysis Plan

4.2.5 **Missing Data** 

In case of partially missing date of birth or date of diagnosis, the following rule will be applied: if

year and months are known but day is missing, then the day will be imputed as 15th; in case of only

year known, the day and month will be imputed as 15th June.

Specific rules for handling for missing efficacy assessments are detailed in section 4.11.1.3.

Methods for handling missing concomitant medication and adverse events dates are detailed in

sections 4.8 and 3.2.3.2 respectively.

Imputations will be used to derive parameters, in listings original data will be presented as

collected.

4.2.6 Data Listing

All original and derived parameters will be listed.

All listings will include scheduled and unscheduled measurements.

Unless specified otherwise, data in listings will be presented by Study Part (Part 1 and Part 2),

Cohort (dose group in Part 1), patient, and visit (ordered by date and time within patient).

All listings will display the same number of decimals as in the source data. All raw data will be

reported exactly as provided.

The data for the patients who consented but for any reason did not receive any dose of study drug

(including screening failures) will be also listed but with a label of '\*'and a footnote to flag these.

Populations used to produce listings are defined in section 4.5.

**Tables and Descriptive Statistics** 

Unless specified otherwise summary tables and figures will be presented by Study Part (Part 1 and

Part 2), Cohort (dose group in Part 1) and visit (as applicable); also, overall summaries will be

shown for the two study parts and for all patients pooled together. In general, summary tables will

be structured in three panels: first panel will summarize overall results obtained in the study parts

Symphogen A/S Sym015-01

Statistical Analysis Plan

and in all patients pooled together; second panel will display all dose groups within the Study Part

1; third panel will display all cohorts within the Study Part 2. Changes from baseline in categorical

data may be summarized using shift tables where appropriate; in shift table each study Part and

Cohort will be appear in a different panel, i.e. first panel will be for 'Overall Part 1 + Part 2',

second panel will be for 'Overall Part 1', third panel will be for 'Overall Part 2', then a panel for

each dose groups within Part 1, finally a panel for each cohort within Part 2.

In general, for variables showing multiple possible categories, these will be displayed following

the within variable logic criteria, for example: ECOG categories will be displayed from 0 and

going to grow; where such a logic criterium does not exist (example: gender, ethnicity, SOC, PT),

categories will be displayed by descending frequencies based on the overall all patients pooled

together. In the end, the order used to show categories within variables should be the same in the

three parts of each table.

Unless otherwise stated, continuous data will be summarized using descriptive statistics including:

number of non-missing observations (n), arithmetic mean, standard deviation (SD), median,

minimum, and maximum.

Categorical data will be summarized in terms of the number of patients providing data at the

relevant time point, frequency counts and percentages. Any planned collapsing of categories will

be detailed in the SAP text and the data displays. Unless otherwise specified, percentages will be

calculated using number of patients providing data at the relevant time point as the denominator.

For visits at which less than 10 patients in the expansion cohorts remain on study treatment,

statistical summaries will no longer be produced.

The following rules will apply to all descriptive statistic displays, except the PK concentrations,

and parameters that are reported in significant digits as described below, where 'd' denotes the

decimal places in the original reported value:

n: 0 decimal places (d.p.)

Mean: d + 1 d.p.

TP-GDO-WW-133-01

Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 CONFIDENTIAL


Project Document Effective Date: 05Jun2019


Symphogen A/S Sym015-01

Statistical Analysis Plan

Confidence Interval: d + 1 d.p.

• SD: d + 2 d.p.

Median: d + 1 d.p..

Minimum: d.

Maximum: d.

Statistics in percentage: 1 d.p.

p-value: 4 d.p.

• Except for p-value, a maximum of 3 decimal places will be displayed.

P-values greater than or equal to 0.001, in general, will be presented to three decimal places. P-values less than 0.001 will be presented as "<0.001".

Details for reporting of statistical summaries specific to PK are detailed in section 4.11.4.4.

All tables, listings, and graphs will be produced to landscape orientation using Courier New 9pt font and will be incorporated into a MS Word document as a (RTF) rich text file (margins on standard A4: Margins (top, left, right, and bottom) 2.54 cm.

4.2.8 Figures

If not otherwise specified, each figure will be presented separately for the two study parts with differentiate legend to discriminate the dose groups within the regimen, e.g. different line types can be used for each group; moreover, an overall figure will also be presented with differentiate legend to discriminate the two study parts. In the end, there will be three panel for each figure: first panel will show all patients, second panel patients in study part 1, third panel patients in study part 1.

All figures will be produced in black and white.

Symphogen A/S Sym015-01

Statistical Analysis Plan

4.3 Software

The tables, listings, figures and any non-descriptive statistical analysis will be produced using

SAS® Software (Version 9.3 or higher). The REPORT procedure (SAS PROC Report) will be

used to produce all tables and listings; SAS/GRAPH will be used to produce all figures.

4.4 Study Patients

4.4.1 Disposition of Patients

The patient disposition including the date the informed consent was signed, date of last infusion

of study drug and the primary reason for End of Treatment will be listed. Moreover, the number

of patients who consented to the study, were exposed to study treatment and primary reason for

end of treatment will be summarized.

Those patients who did not meet the eligibility criteria or were screen failures will be listed.

A listing of patients included into each of the analysis set will be presented, related summary

statistics will be provided.

A clear accounting of the disposition of all patients who enter the study will be provided, from

screening to study completion.

4.4.2 Protocol Deviations

A protocol deviation is any change, divergence, or departure from the study design or procedures

of a study protocol. All protocol deviations will be listed by patient. All protocol deviations will

be discussed during Data Review Meeting (DRM) and addressed with the "final" classification

together their overall effect on a patient, as well, assignment of each patient to the analysis sets

will be decided. During DRM, all protocol deviations and their possible impacts will be discussed

between and the Sponsor and will be assessed as "minor" or "major". Major protocol

deviations and protocol deviations affecting primary analyses can lead to the exclusion of a patient

from the analysis sets. Reasons for excluding patients from any analysis set will be reported and

described in the DRM Report that will be finalized before database hard lock and signed off by all

relevant scientific experts.

Symphogen A/S Sym015-01

Statistical Analysis Plan

4.5 Analysis Sets

Analysis sets are defined in accordance with the consolidated ICH E9 GCP guidelines.

The Full Analysis Set (FAS) will comprise all enrolled patients who have received at least one dose of Sym015. The FAS will be used for evaluation of all endpoints except evaluation of DLTs.

The patients in the FAS will contribute to the analyses as allocated to treatment. For the evaluation

of PK endpoints; patients, full profiles, or single measurements can be excluded from the analyses.

The decision of excluding patients, full profiles, or part of profiles will be described in the clinical

trial report (CTR).

The DLT Analysis Set will comprise all patients in the FAS enrolled in Part 1, except patients who

did not complete Cycle 1 (i.e., the initial 28-day period of Q2W dosing) for reasons other than

drug toxicity. The DLT Analysis Set will be used for evaluation of DLTs.

Demographic and Baseline Characteristics and Safety variables will be listed based on all

consented patients, not treated patients will be flagged as specified in section 4.2.6.

Efficacy, Immunology, Pharmacodynamic and Pharmacokinetic variables will be listed based on

FAS.

In general, all summary tables will be produced based on FAS.

DLT listing and DLT event evaluation will be based on DLT Analysis Set.

4.6 Demographics and Baseline Characteristics, Disease History and Prior Cancer

**Therapies** 

The following demographic and baseline variables will be recorded:

Date of informed consent

Date of Birth

Gender, Race and Ethnicity

Height

- · Weight at screening and baseline
- Stage at initial diagnosis and current stage
- Screening and baseline ECOG PS (categories)
- · Disease history and diagnosis, including:
  - Site of primary tumor
  - o Date of initial diagnosis
  - o Histopathologic diagnosis
  - Sites of metastases
  - o MET-amplification Status: Amplified [yes, no, unknown]
  - o Fluorescence In Situ Hybridization (FISH)
  - o Chromogenic In Situ Hybridization (CISH)
  - Silver In Situ Hybridization (SISH)
  - Next-Generation Sequencing (NGS)
  - Quantitative PCR (qPCR)
  - KRAS Mutation Status [Wild Type, Mutated]
  - METex14 Mutation Status [Yes, No, Not Applicable] (only collected from Protocol version 7)
  - o Debulking surgery performed [yes, no], if yes date of debulking
  - Date of most recent progression
- Prior cancer therapies (surgical procedure and prior radiation and systemic therapy including dates of the treatments and, as applicable, body site or location, dose, best

response, reason for discontinuation and progression date).

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 CONFIDENTIAL

Project Document Effective Date: 05Jun2019


Symphogen A/S Sym015-01

Statistical Analysis Plan

Age at consent in years will be derived as (Year of informed consent signed - Year of date of birth)

+ 0 if the month and day of informed consent signed >= the month and day of date of birth, else +

1. The following age classes will be as well derived: < 65 years; 65 - <75 years; 75 - <85 years;

85 years or older.

BMI at baseline will be calculated as Weight [kg] / (Height [m])<sup>2</sup>

Time since initial diagnosis will be derived as (Year of informed consent signed - Year of initial

diagnosis) + 0 if the month and day of informed consent signed >= the month and day of initial

diagnosis, else + 1.

Number of sites with metastases will be derived by counting all sites with metastases.

Prior systemic therapies for cancer will be counted by patient and summarized as 0, 1, 2, 3, 4+ for

each patient.

Regimens containing MET targeting, EGFR targeting, as well as PD1/PDL1 targeting agents will

be manually identified and flagged in the list of the prior systemic therapies.

Anatomic based cancer type categorization will be manually defined for each patient based on

primary tumor site which may also be combined with tumor histology.

Demographic and baseline characteristics, Disease History and Prior Cancer Therapies will be

listed.

Descriptive continuous statistics will be presented for:

· Demographic and baseline characteristics (including age in years, height, weight and

baseline BMI)

Disease History information (including Time since initial diagnosis [years]).


Cancer Gene Mutation as part of Disease History (including FISH, CISH, SISH, NGS and

Quantitative PCR)

The frequency and percentage of patients will be tabulated for:

Symphogen A/S Sym015-01

Statistical Analysis Plan

Demographic and baseline characteristics categorical variables (including age classes,

gender, race, and ethnicity);

Disease History information includes Cancer Baseline Characteristics (Site of primary

tumor, Histopathologic Diagnosis, Anatomic based cancer type, prior debulking surgery

[yes, no], sites of metastases and number of sites with metastasis, baseline ECOG PS) and

Cancer Gene Mutation -(MET amplification Status [Amplified, Non-Amplified], KRAS

Mutation Status [Wild Type, Mutated], METex14 Mutation Status [Yes, No, Not

Applicable]);

• Prior Cancer Therapies (including prior surgical treatment [yes/no], prior radiation therapy

[yes/no], number of prior systemic therapies [0, 1, 2, 3, More than 3]), Prior MET targeting

therapies [yes/no], Prior EGFR targeting therapies [yes/no], Prior PD1/PDL1 targeting

therapies [yes/no].

Date of informed consent, date of birth, weight at screening, Stage at initial diagnosis and current

stage, ECOG at screening, date of initial diagnosis and date of most recent progression will only

be listed.

4.7 Medical History

Medical history is assessed at screening and include prior and ongoing medical illnesses and

conditions and prior surgical procedures not related to the primary diagnosis.

Medical History terms will be coded using Medical Dictionary for Regulatory Activities

(MedDRA) version 22.0 or later version. Medical History terms will be listed only.

4.8 Prior and Concomitant Medications and Concomitant Procedures

Medications are all prescription medications, over-the-counter medications, or alternative

therapies registered from screening through 30 days after the last dose of study drug. Medications

will be listed (excluding Premedication for Sym015 Infusions which will be listed separately).

TP-GDO-WW-133-01 Effective Date: 05 Sep 18

Related to: SOP-GDO-WW-019

CONFIDENTIAL Project Document Version No. 1.0
Project Document Effective Date: 05Jun2019


Symphogen A/S Sym015-01

Statistical Analysis Plan

Medications will be coded using the World Health Organization Drug Dictionary (WHODD),

version global 2019 March B3 or later version and will be presented by WHODD Anatomical-

Therapeutic-Chemical (ATC) therapeutic classification and preferred term (PT).

Medications and treatments administered prior to the first infusion of study drug which stopped

prior to first infusion of study drug will be considered as prior medications and flagged in the

listing.

Medications and treatments which started before, on or after the first infusion of study drug and

which stopped after first infusion of study drug (including medications and treatments which

stopped the day of first infusion) will be considered as concomitant medications.

If medication start and/or stop dates are missing or partial, the dates will be compared as far as

possible with the date of first dose of study medication. Medications will be assumed to be

concomitant, unless there is clear evidence (through comparison of partial dates) to suggest that

the medication stopped prior to the first dose of study medication. If there is clear evidence to

suggest that the medication stopped prior to the first dose of study medication, the medication will

be assumed to be Prior.

Concomitant procedures performed during the study will be collected and listed.

4.9 Pre-medications for Sym015

A premedication schedule is implemented for all patients treated.

For Part 1 of the trial, premedication is mandatory prior to each dose of Sym015.

For Part 2 of the trial, premedication is mandatory prior to each dose of Sym015 during Cycle 1;

if a patient is without evidence of IRRs after Cycle 1, the Investigator may opt to withdraw

premedication on a patient-by-patient basis with subsequent dosing.

All pre-medications will be listed. Study drug administrations proceeded by premedication will be

flagged in the corresponding listing.

## 4.10 Treatment Exposure and Compliance

Data of study drug infusion including dose reduction and interruption information, patient drug administration irregularities (dose reduction and interruption) and infusion related reaction will be listed.

Duration of the Sym015 exposure, treatment duration, actual number of doses, planned total dose, actual total dose and Relative Dose Intensity (RDI) will be derived as follow:

- Duration of exposure (days) = (last dose date first dose date + 1)
- Actual Treatment duration (days) = (last dose date first dose date + 14)
- Actual Treatment duration (weeks) = (last dose date first dose date + 14) / 7

  Actual Treatment duration (week) will be presented at one decimal place precision.
- Number of treatment cycles initiated (i.e. at least one infusion for the cycle)
- Number of treatment cycles completed (i.e. all cycle infusions were received by the patient)
- Planned total number of doses = (Date of last dose Date of first dose + 1) / 14 rounded
   up to integer
- Planned total dose = Planned dose \* Actual total number of doses received
- Planned treatment duration (weeks) = Actual total number of doses × 2
- Planned treatment duration (days) = Actual total number of doses × 14
- Relative dose intensity (RDI)

RDI (%) =  $100 \times \frac{\text{Sum of all received dose/Actual treatment duration (days)}}{\text{Total planned dose / Planned treatment duration (days)}}$ 

whereas the total planned dose (mg/kg) and planned dose duration are calculated based on the number of doses of the study medication a patient had received at the initially planned dose (mg/kg) for the cycle according to the planned dosing schedule. Example, if a patient received 8 bi-weekly (i.e. dose regimen Q2W) doses of a study medication with a loading dose of 12 mg/kg and rest 9 mg/kg, with 1 dose reduction from 9 mg/kg to 6 mg/kg starting at week 14 and 1 week delay and at week 16, then

RDI (%) = 
$$100 \times \frac{(12+5\times9+2\times6)/119}{(12+7\times9)/112} = 86.6\%$$

The number of initiated and completed cycles of taking Sym015 will be summarized both as categoric (0, 1, 2, 3, 4, 5, 6, >6) and continuous parameter.

Duration of the Sym015 exposure, treatment duration, actual number of doses will be summarized as continuous variables. RDI will be summarized both as categoric (> 100%; 90 % - 100%; 80 % - 90%; 70 % - 80%) and continuous parameter. Swimmer Plot will be presented showing Treatment Duration together with Tumor Response data.

Number of patients who had dose reduction (Any, 1, 2, 3+ times) and dose interruption (Any, 1, 2, 3+ times) will be summarized.

In this section, percentages are intended to be calculated using the number of patients dosed in each group, or the Full Analysis Set for the overall study group, as denominator.

## 4.11 Efficacy Evaluation

### 4.11.1 Analysis and Data Conventions

No formal testing of hypotheses has been planned in this study. Therefore, no formal sample size calculations were performed.

#### 4.11.1.1 Multi-center Studies

There will not be any adjustment for study centers, subgroup analysis based on study centers are not planned.


Symphogen A/S Sym015-01

Statistical Analysis Plan

4.11.1.2 Adjustments for Covariates

No statistical models will be provided for the analysis of Study Endpoints. All study analyses will

be descriptive and will be seen from an exploratory perspective. No adjustment for covariates is

expected.

4.11.1.3 Handling of Dropouts or Missing Data

Efficacy data that are reported as missing will be excluded from all descriptive and non-descriptive

data analysis. There will be no imputation of missing efficacy data.

For general rules about handling of missing data refer to section 4.2.

4.11.1.4 Multiple Comparisons/Multiplicity

Not Applicable.

4.11.1.5 Interim Analyses

No interim analysis is planned other than evaluations for dose escalations. No statistical

adjustments will be made for the interim look of the data during the study.

All relevant safety and toxicity data will be reviewed on an ongoing basis throughout the trial.

4.11.1.6 Examination of Subgroups

Anatomic based cancer type will be used as a subgroup to summarize some study endpoints or as

stratification factor in certain graphics as appropriately described in the text of this SAP. Anatomic

based cancer type categorization is derived as described in section 4.6.

4.11.2 Analysis of Efficacy Variable

All statistical analysis of the efficacy endpoints will be presented using the FAS.

All Efficacy Endpoints will be listed.

Time to Event endpoints (TTP, PFS, OS) will be listed at 1 d.p. precision.

Symphogen A/S Sym015-01

Statistical Analysis Plan

In this section, percentages are intended to be calculated using the number of patients dosed in

each group, or the Full Analysis Set for the overall study group, as denominator.

4.11.2.1 Anti-Tumor Response according to RECIST v1.1

The following anti-tumor response endpoints will be measured:

• Number and percentage of patients with documented confirmed OR will be summarized

by Study Part and Cohort (dose group in Part 1) using frequency distribution with the

corresponding 90% exact Clopper-Pearson Confidence Intervals (CI) for binomial

proportion. All documented confirmed ORs will be listed.

• Duration of response (DR) will be listed and summarized as a continuous variable by Study

Part and Cohorts (dose group in Part1)

• Best overall response (BOR) will be listed and summarized by Study Part and Cohorts

(dose group in Part1) using frequency distribution for the categories

Confirmed/Unconfirmed CR, Confirmed/Unconfirmed PR, SD, PD, and Not Evaluable.

Patients in DCR will be listed and summarized by Study Part and Cohorts (dose group in

Part1) using frequency distribution with the corresponding 90% exact Clopper-Pearson

Confidence Intervals (CI) for binomial proportion.

Stable Disease (SD)

Number and percentage of patients with SD duration  $\geq 4$  months and SD  $\geq 6$  months will

be presented summarized by Study Part and Cohorts (dose group in Part1).

Changes in sum of diameters of target lesions from baseline

Changes in the sum of diameters of target lesions from baseline will be listed as percentage

and absolute value, the best change (i.e. the nadir, largest reduction or smallest increase)

will be identified and presented using summary table and plotted with a waterfall plot.

Change in sum of diameters will also be presented by anatomic based cancer type.


Symphogen A/S Sym015-01

Statistical Analysis Plan

Time to Progression (TTP)

TTP will be analyzed with Kaplan Meier product-limit method. The median TTP, as well

as 6-month and 12-month progression rates and the corresponding 90% CIs will be

estimated using the product-limit method and presented using a Kaplan-Meier plot with

median TTP rate marked, and the number of patients at-risk presented at 2, 4, 6, 8, 10 and

12 months, and each two months going forward, as applicable.

Progression Free Survival (PFS)

PFS, including PFS per additional sensitivity analysis, will be analyzed with Kaplan Meier

product-limit method. The median PFS, as well as 6-month and 12-month progression rates

and the corresponding 90% CIs will be estimated using the product-limit method and

presented using a Kaplan-Meier plot with median PFS rate marked, and the number of

patients at-risk presented at 2, 4, 6, 8, 10 and 12 months, and each two months going

forward, as applicable.

Overall Survival (OS)

OS will be analyzed with Kaplan Meier product-limit method. The median OS, as well as

6-month and 12-month progression rates and the corresponding 90% CIs will be estimated

using the product-limit method and presented using a Kaplan-Meier plot with median OS

rate marked, and the number of patients at-risk presented at 6, 12, 18, and 24 months, and

each six months going forward, as applicable.

Results of the tumor evaluation by CT/MRI for target lesions, non-target lesions and tumor

response will be listed.

4.11.3 Pharmacodynamic and Immunogenicity

These variables include:

Tumor markers: Evaluated at timepoints coinciding with the CT/MRI imaging studies

Archival Tumor Tissue for MET and KRAS

Symphogen A/S Sym015-01

Statistical Analysis Plan

Tumor Biopsy for MET Status

Tumor Biopsy for Eligibility and Biomarkers Analysis

Blood Sample for Genomic and Biomarker Analyses. Potential biomarkers of interest

include genes, gene transcripts and proteins of the RTKs and molecules of the MET

signalling pathway, including MET, HGF, EGFR, HER2, HER3, IGF1R, ROS1, RET,

PIK3CA, PTEN, cMYC, KRAS, NRAS, BRAF, AKT1, FGFR, and RON. Analysis of

biomarker blood samples may include genes and/or proteins that are unknown or have not

been included in the scientific hypotheses of this trial, but that, during the collection of data

from this trial, may evolve as new candidate genes and markers related to Sym015 safety,

efficacy, or mechanism of action.

Skin Biopsy results (Part 1 only).

Anti-drug antibody (ADA) Testing.

All these data will be listed.

Data driven exploratory analysis may be conducted according to the study exploratory objectives

based on the available Pharmacodynamic data.

Percentage and nominal change in target expression (parameters) from baseline to end of Cycle 2

or PD (whichever comes first) in skin biopsy samples will be presented in study part 1.

Descriptive statistics will be used, including scatter plots of values at end of Cycle 2 versus

baseline.

4.11.4 Pharmacokinetics

4.11.4.1 Pharmacokinetic Concentrations

The serum concentration of Sym015 is defined as the sum of the serum concentration of the

constituent antibodies, Hu9006 and Hu9338. Serum concentrations for Sym015 and each of the

constituent antibodies, Hu9006 and Hu9338 will be listed by Study Part, cohort (dose group in

Part 1), patient, including actual time relative to dosing (minutes), scheduled time (derived based

Symphogen A/S Sym015-01

Statistical Analysis Plan

on datetime of dosing and schedule of PK assessments) and time deviation from scheduled time

(minutes).

The following definitions are used for PK plots and tables:

• First profile: all PK data points from Cycle 1 Day 1 to Cycle 1 Day 15 (pre-dose)

Dosing/sampling occasions: Week 1, 3, 5, 7, 9 etc., EOT, 1MFUP

Peaks: serum concentration assessed at EOI for each dosing occasion

Troughs: serum concentrations assessed prior to SOI for each dosing occasion

Violations of scheduled sampling will be reviewed on a patient by patient basis by Symphogen and Following data review by Symphogen's pharmacokinetic expert, data points may

be excluded from mean calculations and parameter calculation based on the below criteria:

Individual outlying data points which are markedly deviating from the preceding and

following time points

Data points or PK profiles which are not compatible with known physiological processes

underlying the PK properties

• Unexpected events or protocol deviations documented in e.g. laboratory notes or in

protocol deviation reviews

Exclusions will be documented in the study files and the PC/PP files.

Patient profiles of Sym015 plasma concentrations vs. time points will be plotted by Study Part and

cohort (dose group in Part 1) and analyte (Hu9006, Hu9038 or Sym015). Following plots will be

produced:

• Patient Profiles (one panel for each patient) with overlays of Sym015, Hu9006, and

Hu9038 concentration vs. actual time by Study Part and Cohort (First profile) – Linear

Patient Profiles (one panel for each patient) with overlays of Sym015, Hu9006, and

Hu9038 concentration vs. actual time by Study Part and Cohort (First profiles) - Semi-log

TP-GDO-WW-133-01

Effective Date: 05 Sep 18

Related to: SOP-GDO-WW-019


Project Document Effective Date: 05Jun2019


 Patient Profiles (one panel for each patient) with overlay of Sym015, Hu9006, and Hu9038 concentration vs. actual time by Study Part and Cohort (peak and trough for each dosing occasion) – Linear

 Patient Profiles (one panel for each patient) with overlay of Sym015, Hu9006, and Hu9038 concentration vs. actual time by Study Part and Cohort (peak and trough for each dosing occasion) – Semi-log

Descriptive summary (n, arithmetic mean, SD, median, minimum, maximum, geometric means, and geometric CV%) of serum concentrations of Sym015, Hu9006, and Hu9038 and fraction Hu9006 (concentration of Hu9006/concentration of Sym015) will be tabulated by dose schedule, dose group and nominal sampling time. Following tables will be produced:

- Summary of Sym015, Hu9006, and Hu9038 concentration, and fraction Hu9006 by Cohort and Time Point (First profile)
- Summary of Sym015, Hu9006, and Hu9038 concentration, and fraction Hu9006 by Cohort and Time Point (Peak and trough for each dosing occasion)

The arithmetic and geometric means of the plasma concentrations of Sym015 vs. nominal time points will be plotted by dose group with +/-1 standard deviation (for arithmetic means). In figures of geometric means, error bars will be calculated using the following formula: Exp (mean\_Ln +/-sd\_Ln) where 'sd\_Ln' denotes the standard deviation of the concentration values on the log base 10 scale and 'mean\_Ln' denotes the arithmetic mean of the concentration values on the log base 10 scale. The following mean concentration vs. time plots will be produced for each analyte (Sym015, Hu9006 and Hu9038):

- Arithmetic Mean Concentration of <Analyte> vs. planned time point by cohort (First profile) Linear
- Geometric Mean Concentration of <Analyte> vs. planned time point by cohort (First profile) Semi-log
- Arithmetic Mean Peak and Trough Concentrations of <Analyte> vs. planned time point by cohort (peaks and troughs at all dosing occasions) – Linear

Symphogen A/S Sym015-01

Statistical Analysis Plan

• Geometric Mean Peak and Trough Concentrations of <Analyte> vs. planned time point

by cohort (peaks and troughs at all dosing occasions) - Semi-log

4.11.4.2 Handling of Values Below the Limit of Quantification (BLO)

In summary tables, values below the LLOQ (BLQ) will be handled as follows:

• At a time point where less than or equal to 50% of the values are BLQ, all BLQ values will

be set to the ½\*lower limit of quantification (LLOQ), and all descriptive statistics will be

calculated.

• At a time point where more than 50% of the values are BLQ, the mean, SD, geometric

mean and CV% will be set to Not Determined (ND). The max value will be reported from

the individual data, and the min and median will be set to BLQ.

• If all values are BLQ at a time point, no descriptive statistics will be calculated for that

time point. Not Applicable (NA) will be written in the field for SD and CV% and BLQ will

be written in fields for mean, geometric mean, min, median, and max.

The number of BLQ values (n below LLOQ) will be reported for each time point.

In figures, all BLQ values will be set to the ½\*LLOQ.

4.11.4.3 Pharmacokinetic Parameters

Pharmacokinetic parameters for the first profile for each patient and analyte (Sym015, Hu9006,

Hu9038) will be derived by model-independent, non-compartmental analysis (NCA) according to

Symphogen's local procedures.

All derived serum PK parameters will be listed by Study Part and Cohort (dose group in Part 1),

patient, and Day, and summarized descriptively by Study Part and Cohort (dose group in Part 1)

and Day. The following descriptive statistics will be presented for PK parameters: n, arithmetic

mean, SD, geometric mean, geometric CV% (calculated as: gCV%=SQRT(exp(s²)-1)\*100; where

s is the standard deviation of the log-transformed values), median, minimum and maximum values.


## 4.11.4.4 Pharmacokinetic Analysis

Descriptive statistics of plasma concentrations will be reported with the same precision as the source data and plasma concentrations.

In addition to general continuous summary statistics presented in section 4.2, for PK parameters, geometric means with coefficient of variation (CV %) will be also summarized.

For drug concentrations and concentration-dependent pharmacokinetic parameters, the rules of data presentation are described in table below.

## Presentation of PK Parameters and Summary Statistics

| Typical<br>Variable | N | Digit rule | Minimum/<br>Maximum | Mean<br>Median | SD | Geometric<br>Mean | CV<br>(%) |
|---|---|---|---|---|---|---|---|
| concentration | X | Significant digits | 3 | 4 | 4 | 3 | 3 |
| $C_{\text{max}}$ | X | Significant digits | 3 | 4 | 4 | 4 | 4 |
| $t_{max}^{*}$ | X | Fixed decimal places | as raw data | as raw data | <b>3</b> | ÷ | <u>a</u> |
| $\lambda_z$ | X | Significant digits | 4 | 3 | 5 | 5 | 5 |
| t <sub>1/2</sub> | X | Significant digits | 3 | 3 | 4 | 4 | 4 |
| AUC <sub>(0-xx)</sub> | X | Significant digits | 3 | 3 | 4 | 4 | 4 |
| $\mathrm{AUC}_{(0-\tau)}$ | X | Significant digits | 3 | 3 | 4 | 4 | 4 |

<sup>\*</sup> Mean and SD, geometric mean and CV will not be calculated for t<sub>max</sub>.

# 4.12 Safety Evaluation

### 4.12.1 Dose Limiting Toxicities (DLT)

All DLT events occurred in Cycle 1 will be listed in DLT analysis set. Presence and absence of DLTs will be presented for patients in DLT analysis set.

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 CONFIDENTIAL


Symphogen A/S Sym015-01

Statistical Analysis Plan

4.12.2 Adverse Events

The AEs will be coded using MedDRA version22.0 or later version.

In AE summary tables, percentages will be calculated using the number of patients dosed in each

group, or the Full Analysis Set for the overall study group, as denominator.

TEAEs will be presented by MedDRA System Organ Class (SOC) and Preferred Term (PT). In all

AE summary tables, SOCs and PTs will be presented in the order of descending frequencies as

detailed in section 4.2. AE frequency accounts for number and percent of patients who have a

specific SOC and PT as well as the worst grade, if there were multiple occurrences at different

toxicity grade, which was determined using CTCAE v4.03.

For purposes of the summary tables, AEs will be classified as either being related to study drug or

not related. AEs related to study drug will include AEs classified as 'Related', 'Probably Related'

or 'Possibly Related'. AEs not related to study drug will include AEs that are 'Unlikely Related'

or 'Not Related'.

All AEs will be listed. The AEs will be presented using summary tables including:

• Patient Overall Summary of TEAEs. This table will include following summaries:

o Any TEAEs

Any related TEAEs

Any Serious TEAEs

o Any related Serious TEAEs

Grade 3 or higher TEAEs

Any Related Grade 3 or higher TEAEs

Any TEAEs leading to Permanent Discontinuation of IMP

Any Related TEAEs leading to Permanent Discontinuation of IMP

Related to: SOP-GDO-WW-019


- Any TEAEs leading to interruption or Stop of study drug
- Any Related TEAEs leading to interruption or Stop of study drug
- Any TEAEs with an outcome of reduction or delay of study drug
- o Any Relate TEAEs with an outcome of reduction or delay of study drug
- Any FATAL TEAEs
  - Fatal TEAEs within 30 days from last IMP infusion
  - Fatal TEAEs at more than 30 days from last IMP infusion
- TEAEs by SOC and PT
- Related TEAEs by SOC and PT
- TEAEs by SOC and PT and Worst CTCAE Grade
- Related TEAEs by SOC and PT and Worst CTCAE Grade
- Serious TEAEs by SOC and PT
- Related Serious TEAEs by SOC and PT
- TEAEs Leading to Permanent Discontinuation of IMP by SOC and PT
- Related TEAEs Leading to Permanent Discontinuation of IMP by SOC and PT
- Serious Adverse Events Key Patient Information
- Adverse Events with Outcome of Death Key Patient Information (non TEAEs will be flagged)
- Adverse Events Leading to Permanent Discontinuation of IMP Key Patient Information
- Adverse Events Leading to Dose Reduction Key Patient Information
- Adverse Events Leading to Dose Interruption or Stop- Key Patient Information

 Listing of Death (Deaths occurring within 30 days from last infusion of IMP will be identified; non TEAEs will be flagged)

Key Patients Information will include Patient number, gender and age, AE SOC, PT and Reported Term, AE Serious (Yes / No), AE start and end date and AE duration (days), AE Relationship to Study Drug, TEAE (Yes / No); additional information may also be reported in different listing.

4.12.3 Deaths, Serious Adverse Events, and Other Significant Adverse Events

Reporting of Deaths, Serious Adverse Events and other significant Adverse Events is described in the above section 4.12.2.

4.12.4 Clinical Laboratory Evaluation

All clinical laboratory test results will be presented and summarized using the International System of Units (SI units; Système International d'Unités). The original lab test units will be converted to SI according to Young, D.S and Huth, E.J; 1998; SI Units for Clinical Measurement; American College of Physicians; Philadelphia and Burtis, C.A, Ashwood, E.R and Bruns, D.E; 2008; Fundamentals of Clinical Chemistry; Saunders Elsevier; Missouri [Laboratory test converted to SI will be stored in SDTM LB domain as LBSTRESU and LBSTRESC].

Descriptive statistics (n, mean, standard deviation, median, and range) of the lab parameters and changes from baseline will be presented in SI units for biochemistry, hematology, and coagulation. Such descriptive statistics will be presented by Visit and at End of Study; by Visit summaries will be presented based on worst by-visit result as detailed in section 4.12.4. Worst Result during Treatment (i.e. Maximum and Minimum observed result post Baseline and corresponding change from baseline including results from unscheduled and repeated assessments) will be presented as well.

Shift in biochemistry, hematology, and coagulation result CTCAE grading from baseline to visit maximal grade will be tabulated by each visit and at the end of treatment, as well as from baseline to the maximal grade during the whole study (maximal grade will also include results from unscheduled and repeated assessments).

Symphogen A/S Sym015-01

Statistical Analysis Plan

All clinical laboratory test results will be listed in the original and SI units, for biochemistry,

hematology, coagulation, and urinalysis. Listing of abnormal values will be provided as well.

Individual patient biochemistry, hematology, and coagulation parameters during the trial can be

presented graphically using longitudinal spaghetti plots. Specific lab parameters to be plotted will

be decided by Symphogen from clinical meaning perspective after examination of corresponding

listings.

Selected biochemistry, hematology, and coagulation parameters will be presented using box plots

by visits and Anatomic based cancer type. Specific lab parameters to be plotted will be decided by

Symphogen from clinical meaning perspective after examination of corresponding listings.

Results from the pregnancy tests will be listed.

4.12.5 Echocardiogram (ECHO) or Multi-Gated (MUGA) Scan

ECHO/MUGA data will be listed.

4.12.6 Vital Signs

Data for vital signs (weight, blood pressure, heart rate, temperature) will be listed.

Descriptive summary statistics (for observed values and changes from baseline) for vital sign

parameters will be provided.

4.12.7 Electrocardiograms (ECG)

ECG parameter data will be listed.

Normal, abnormal, or abnormal clinically significant ECG will be presented in a summary table.

A shift from baseline table will be presented as well. Number and percentage of patients with

maximum postdose QTcF values of <=450, >450 ms and <=480, >480 ms and <=500, and >500

ms, and maximal change from baseline values of <=30, >30 and <=60ms, and >60 ms will be at

each scheduled timepoint as well as the highest measurement during the study and at end of

treatment. (highest QTcF Prolongations measurement will also include results from unscheduled

and repeated assessments). Above categories of QTcF are based on ICH E14 [9].


Symphogen A/S Sym015-01

Statistical Analysis Plan

4.12.8 Physical Examination

All results from the physical examination will be listed.

Normal, abnormal not clinically significant, or abnormal clinically significant physical

examination will be summarized by Body System. A shift table from baseline of normal and

abnormal findings in physical examination will be presented.

4.12.9 Eastern Cooperative of Oncology Group (ECOG) Performance Status (PS)

ECOG performance status will be listed.

Number of patients reporting each ECOG score will be presented; a shift table will also be

presented to show changes from Baseline.

4.13 Safety Monitoring

A safety monitoring committee (SMC) is established and includes Investigator(s), Medical

Monitor(s), and Sponsor's medical representatives. The SMC reviewed clinical and laboratory

safety data regularly throughout the trial. The SMC selected the Q2W RP2D to be used in Part 2

based on safety data and available PK results.

The annual Development Safety Update Report (DSUR) was submitted by the Sponsor or designee

to all appropriate Health Authorities and central IRBs/ECs as per ICH Guidelines. Submission of

the DSUR to local IRBs/ECs was handled as per local regulations and/or requests.

4.14 Other Analyses

No other analyses planned.

4.15 Determination of Sample Size

The primary endpoint of Part 1 of the trial is the occurrence of DLTs measured during Cycle 1 of

Sym015 administration. The number of enrolled patients will depend on the extent of observed

DLTs independently in each cohort. Based on a 3+3 design, it is planned to enroll between 12 and

15 patients during dose-escalation, however the actual number of patients will depend on observed

DLTs.

Symphogen A/S Sym015-01

Statistical Analysis Plan

In Part 2 of the trial, the primary endpoint is documented, confirmed OR assessed by RECIST

v1.1, at any time during trial participation by Investigator assessment. It is planned to include 25

patients with various advanced solid tumor malignancies, documented and confirmed as MET-

amplified in the Basket Cohort, 20 patients in the NSCLC MET-Amplified Cohort, and 6-12

patients in the NSCLC MET<sup>Ex14Del</sup> Cohort, for the total of approximately 51-57 patients in Part 2.

No power and type I error considerations were used to determine the sample size in each cohort.

Proposed sample sizes in Basket and NSCLC Cohorts should allow to obtain preliminary safety,

PK, response, and pharmacodynamic information of Sym015 in the respective patient populations.

The expected (target) range of OR in any of these three cohorts is in the range of 20%-50%,

depending on histology, previous therapies, and other prognostic factors defining the enrolled

patient population.

4.16 Changes in the Conduct of the Study or Planned Analysis

DCR analysis was not included as part of study endpoints in the Protocol, such analysis

has been added in this SAP.

• Protocol defines SD for >4 months as a secondary endpoint, this has been changed to SD

for  $\geq$ 4 months, moreover SD for SD for  $\geq$ 6 months has been added as well.

Analysis of Changes in sum of diameters of target lesions from baseline to end of trial

participation was not included as part of study endpoints in the Protocol, such analysis has

been added in this SAP.

Additional sensitivity analysis has been added for PFS as described is sections 3.2.1.1 and

4.11.2.1.

Symphogen A/S Sym015-01

Statistical Analysis Plan

5 REFERENCES

[1] WHO World Cancer Report 2014. Edited by Bernard W. Stewart and Christopher P. Wild.

[2] Dela Cruz CS, Tanoue LT, and Matthay RA. Lung cancer: Epidemiology, etiology, and

prevention. Clin Chest Med 2011; 32(4):doi:10.1016/j.ccm.2011.09.001.

[3] Petrini I: Biology of MET: a double life between normal tissue repair and tumor progression.

Ann Transl Med. 2015 Apr;3(6):82.

[4] Kawakami H, Okamoto I, Okamoto W, et al: Targeting MET Amplification as a New

Oncogenic Driver. Cancers (Basel). 2014 Jul 22;6(3):1540-52.

[5] Sacco JJ, Clague MJ: Dysregulation of the Met pathway in non-small cell lung cancer:

implications for drug targeting and resistance. Transl Lung Cancer Res. 2015 Jun;4(3):242-52.

[6] Eisenhauer EA, Therasse P, Bogaerts J, et al: New response evaluation criteria in solid tumors:

Revised RECIST guideline (version 1.1). Eur J Cancer 2009; 45:228-247.

[7] Clinical Trial Endpoints for the Approval of Cancer Drugs and Biologics, December 2018,

U.S. Department of Health and Human Services Food and Drug Administration Oncology Center

of Excellence.

[8] ICH HARMONISED TRIPARTITE GUIDELINE, STRUCTURE AND CONTENT OF

CLINICAL STUDY REPORTS, E3, 30 November 1995

[9] ICH HARMONISED TRIPARTITE GUIDELINE; THE CLINICAL EVALUATION OF

QT/QTC INTERVAL PROLONGATION AND PROARRHYTHMIC POTENTIAL FOR NON-

ANTIARRHYTHMIC DRUGS; E14.

[10] SAS® Version 9.2 of the SAS System for Personal Computers. Copyright © 2002-2003. SAS

Institute Inc. SAS and all other SAS Institute Inc. product or service names are registered

trademarks or trademarks of SAS Institute Inc., Cary, NC, USA.

#### 6 TABLES, FIGURES and LISTINGS

- Table 14.1.1 Patients Enrollment (All Consented Patients)
- Table 14.1.2 Patient Disposition by Part, Dose Group and Cohort (Full Analysis Set)
- Table 14.1.3 Patient Demographics and Baseline Characteristics (Full Analysis Set)
- Table 14.1.4 Cancer Baseline Characteristics (Full Analysis Set)
- Table 14.1.5 Cancer Gene Mutation (Full Analysis Set)
- Table 14.1.6 Prior Cancer Therapies (Full Analysis Set)
- Table 14.2.1.1 Serum Concentration of Sym015 constituent antibodies, first profile (Full Analysis Set)
- Table 14.2.1.2 Peak and Trough Serum Concentration of Sym015 constituent antibodies by Study Day (Full Analysis Set)
- Table 14.2.1.3 Serum PK Parameters of Sym015 (Full Analysis Set)
- Table 14.2.2 Biomarkers from Skin Biopsy (Full Analysis Set)
- Table 14.2.3.1 Best Overall Response, Objective Response and Disease Control Rate (Full Analysis Set)
- Table 14.2.3.2 Time to Progression, Duration of Stable Disease and Duration of Response (Full Analysis Set)
- Table 14.2.3.3 Progression Free Survival, Overall Survival (Full Analysis Set)
- Table 14.2.3.3 Maximal Reduction in Sum of Diameters of Target Lesion from Baseline (Full Analysis Set)
- Table 14.2.3.4 Maximal Reduction in Sum of Diameters of Target Lesion from Baseline by Anatomic based cancer type (Full Analysis Set)

Table 14.2.3.5 Number of Treatment Cycles (Full Analysis Set)

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 CONFIDENTIAL


- Table 14.2.3.6 Treatment Duration and Dose Intensity (Full Analysis Set)
- Table 14.2.3.7 Dose Reduction, Interruption, and Delay (Full Analysis Set)
- Table 14.2.3.8 Dose-Limiting Toxicity (DLT Analysis Set)
- Table 14.3.1.1 Overall Summary of TEAEs (Full Analysis Set)
- Table 14.3.1.2 TEAEs by SOC and PT (Full Analysis Set)
- Table 14.3.1.3 Related TEAEs by SOC and PT (Full Analysis Set)
- Table 14.3.1.4 TEAEs by SOC and PT and Worst CTCAE Grade (Full Analysis Set)
- Table 14.3.1.5 Related TEAEs by SOC and PT and Worst CTCAE Grade (Full Analysis Set)
- Table 14.3.1.6 Serious TEAEs by SOC and PT (Full Analysis Set)
- Table 14.3.1.7 Related Serious TEAEs by SOC and PT (Full Analysis Set)
- Table 14.3.1.8 TEAEs Leading to Permanent Discontinuation of IMP by SOC and PT (Full Analysis Set)
- Table 14.3.1.9 Related TEAEs Leading to Permanent Discontinuation of IMP by SOC and PT (Full Analysis Set)
- Listing 14.3.2.1 Serious Adverse Events Key Patient Information (Full Analysis Set)
- Listing 14.3.2.2 Adverse Events with Outcome of Death Key Patient Information Full Analysis Set
- Listing 14.3.2.3 Adverse Events Leading to Permanent Discontinuation of Investigational Product Key Patient Information Full Analysis Set
- Listing 14.3.2.4 Adverse Events Leading to Dose Reduction Key Patient Information Full Analysis Set
- Listing 14.3.2.5 Adverse Events Leading to Infusion Interruption or Stop Key Patient Information Full Analysis Set

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Listing 14.3.2.6 Listing of Death (Full Analysis Set)

Listing 14.3.4.1 Abnormal Hematology Values

Listing 14.3.4.2 Abnormal Chemistry and Coagulation Values

Listing 14.3.4.3 Abnormal Urinalysis Values

Table 14.3.5.1 Clinical Laboratory Hematology-Summary of Observed Values and Change from Baseline by Visit (Full Analysis Set)

Table 14.3.5.2 Clinical Laboratory Chemistry-Summary of Observed Values and Change from Baseline by Visit (Full Analysis Set)

Table 14.3.5.3 Clinical Laboratory Coagulation-Summary of Observed Values and Change from Baseline by Visit (Full Analysis Set)

Table 14.3.5.4 Clinical Laboratory Hematology -Summary of CTCAE Grade Shift from Baseline to Maximal Grade (Full Analysis Set)

Table 14.3.5.5 Clinical Laboratory Chemistry – Summary of CTCAE Grade Shift from Baseline to Maximal Grade (Full Analysis Set)

Table 14.3.5.6 Clinical Laboratory Coagulation – Summary of CTCAE Grade Shift from Baseline to Maximal Grade (Full Analysis Set)

Table 14.3.6.1 Vital Signs Observed Values and Change from Baseline by Visit (Full Analysis Set)

Table 14.3.6.2 ECG Clinical Assessment by Visit (Full Analysis Set)

Table 14.3.6.3 ECG Shift from Baseline by Timepoint (Full Analysis Set)

Table 14.3.6.4 ECG- QTcF Prolongations Summary (Full Analysis Set)

Table 14.3.6.5 Physical Examination Clinical Assessment by Visit (Full Analysis Set)

Table 14.3.6.6 Physical Examination Shift from Baseline by Timepoint (Full Analysis Set)

Table 14.3.6.7 ECOG-PS by Visit (Full Analysis Set)

Table 14.3.6.8 ECOG-PS Shift from Baseline by Timepoint (Full Analysis Set)

Figure 14.2.1 Skin Biopsy: scatter plot of values at End of Cycle 2 versus Baseline (Part 1, Full Analysis Set)

Figure 14.2.2 Patient Profiles for all analyte concentration versus Actual Time by Study Part and Cohort – First Profile – Linear (Full Analysis Set)

Figure 14.2.3 Patient Profiles for all analyte concentration versus Actual Time by Study Part and Cohort – First Profile – Semi-log (Full Analysis Set)

Figure 14.2.4 Patient Profiles for all analyte concentration versus Actual Time by Study Part and Cohort – Peak and Trough all dosing occasions – Semi-log (Full Analysis Set)

Figure 14.2.5 Patient Profiles for all analyte concentration versus Actual Time by Study Part and Cohort – Peak and Trough all dosing occasions – Semi-log (Full Analysis Set)

Figure 14.2.6 Arithmetic Mean Concentration of all analyte versus nominal Time Point by Analyte, Study Part and Cohort First Profile – Linear (Full Analysis Set)

Figure 14.2.7 Geometric Mean Concentration of all analyte versus nominal Time Point by Analyte, Study Part and Cohort First Profile – Semi-log (Full Analysis Set)

Figure 14.2.8 Arithmetic Mean Peak and Trough Concentrations of all analyte versus nominal Time Point by Analyte, Study Part and Cohort peaks and troughs at all dosing occasions – Linear (Full Analysis Set)

Figure 14.2.9 Geometric Mean Peak and Trough Concentrations of all analyte versus nominal Time Point by Analyte, Study Part and Cohort peaks and troughs at all dosing occasions – Semilog (Full Analysis Set)

Figure 14.2.10 Spaghetti Plot for Selected Hematology parameters (Full Analysis Set)

Figure 14.2.11 Spaghetti Plot for Selected Biochemistry parameters (Full Analysis Set)

- Figure 14.2.12 Spaghetti Plot for Selected Coagulation parameters (Full Analysis Set)
- Figure 14.2.13 BoxPlot for Selected Hematology parameters by Visit (Full Analysis Set)
- Figure 14.2.14 BoxPlot for Selected Biochemistry parameters by Visit (Full Analysis Set)
- Figure 14.2.15 BoxPlot for Selected Coagulation parameters by Visit (Full Analysis Set)
- Figure 14.2.16 BoxPlot for Selected Hematology parameters by Visit and Anatomic based cancer type (Full Analysis Set)
- Figure 14.2.17 BoxPlot for Selected Biochemistry parameters by Visit and Anatomic based cancer type (Full Analysis Set)
- Figure 14.2.18 BoxPlot for Selected Coagulation parameters by Visit and Anatomic based cancer type (Full Analysis Set)
- Figure 14.2.19 Waterfall Plot of the Best Percent Change from Baseline in Sum of Diameters of Target Lesions (Full Analysis Set)
- Figure 14.2.20 Waterfall Plot of the Best Percent Change from Baseline in Sum of Diameters of Target Lesions by Anatomic based cancer type (Full Analysis Set)
- Figure 14.2.21 Kaplan Meier Survival Curve for Time To Progression (Full Analysis Set)
- Figure 14.2.22 Kaplan Meier Survival Curve for Progression Free Survival (Full Analysis Set)
- Figure 14.2.23 Kaplan Meier Survival Curve for Progression Free Survival Sensitivity Analysis (Full Analysis Set)
- Figure 14.2.24 Kaplan Meier Survival Curve for Overall Survival (Full Analysis Set)
- Figure 14.2.25 Swimmer Plot of Duration of Treatment and Tumor Response (Full Analysis Set)
- Listing 16.2.1.1 Patients Disposition (All Consented Patients)
- Listing 16.2.1.2 Screen Failure and Patients Not Meeting Eligibility Criteria (All Consented Patients)

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019 CONFIDENTIAL.


Symphogen A/S Sym015-01

Statistical Analysis Plan

Listing 16.2.2.1 Protocol Deviations (All Consented Patients)

Listing 16.2.3.1 Analysis Sets (All Consented Patients)

Listing 16.2.4.1 Demographics and Baseline Characteristics (All Consented Patients)

Listing 16.2.4.2 Medical and Surgical History (All Consented Patients)

Listing 16.2.4.3.1 Prior and Concomitant Medications (All Consented Patients)

Listing 16.2.4.3.2 Concomitant Procedures (All Consented Patients)

Listing 16.2.4.3.3 Premedication for Sym015 (All Consented Patients)

Listing 16.2.4.4.1 Cancer Diagnosis (All Consented Patients)

Listing 16.2.4.4.2 Cancer Gene Mutation (All Consented Patients)

Listing 16.2.4.4.3 Prior Cancer Therapies: Surgical Procedure (All Consented Patients)

Listing 16.2.4.4.4 Prior Cancer Therapies: Radiation Therapy (All Consented Patients)

Listing 16.2.4.4.5 Prior Cancer Therapies: Systemic Therapy (All Consented Patients)

Listing 16.2.5.1 Study Drug Administration (Full Analysis Set)

Listing 16.2.5.2 Study Drug Administration Irregularities (Full Analysis Set)

Listing 16.2.5.3 Study Drug Infusion Related Reaction (Full Analysis Set)

Listing 16.2.6.1 Pharmacokinetic Blood Sampling and Serum Concentrations of Sym015 Analytes (Full Analysis Set)

Listing 16.2.6.2 Sym015 Serum PK Parameters (Full Analysis Set)

Listing 16.2.6.3 Pharmacodynamics Parameters - Biomarkers (Full Analysis Set)

Listing 16.2.6.4.1 Tumor Assessment - Target Lesion (Full Analysis Set)

Listing 16.2.6.4.2 Tumor Assessment – Non-Target Lesion (Full Analysis Set)

Symphogen A/S Sym015-01

Statistical Analysis Plan

Listing 16.2.6.4.3 Tumor Response by Visit (Full Analysis Set)

Listing 16.2.6.5 Best Overall Response, Objective Response, Time To Progression, Disease Control Rate (Full Analysis Set)

Listing 16.2.6.6 Progression Free Survival (Full Analysis Set)

Listing 16.2.6.7 Overall Survival (Full Analysis Set)

Listing 16.2.7.1 Dose Limiting Toxicity (DLT Analysis Set)

Listing 16.2.7.2 Adverse Events (All Consented Patients)

Listing 16.2.8.1 Clinical Laboratory Hematology Results and Change from Baseline (All Consented Patients)

Listing 16.2.8.2 Clinical Laboratory Chemistry and Coagulation Results and Change from Baseline (All Consented Patients)

Listing 16.2.8.3 Clinical Laboratory Urinalysis Results (All Consented Patients)

Listing 16.2.8.4 Pregnancy Test (All Consented Patients)

Listing 16.2.9.1 Vital Signs – Observed and Change from Baseline Values (All Consented Patients)

Listing 16.2.9.2 Electrocardiogram (All Consented Patients)

Listing 16.2.9.3 ECHO/MUGA(ECHO) (All Consented Patients)

Listing 16.2.9.4 Physical Examination (All Consented Patients)

Listing 16.2.9.5 ECOG-PS (All Consented Patients)

Symphogen A/S Sym015-01

Statistical Analysis Plan

### 7 APPENDICES

# 7.1 Derivation of CTCAE Grade - Hematological Tests

| Tests | Direction | | Gr | Grade | |
|---|---|---|---|---|---|
| | | | 2 | 3 | 4 |
| Hemoglobin (g/dl, | | <lln -="" 10.0="" 8.0="" <10.0="" dl;="" dl;<="" g="" td=""><td>&lt;10.0 - 8.0 g/dL;</td><td>&lt;8.0 g/dL;</td><td>Life-threatening</td></lln> | <10.0 - 8.0 g/dL; | <8.0 g/dL; | Life-threatening |
| mmol/L | | <lin -="" 6.2<="" td=""><td>&lt;6.2 - 4.9 mmol/L;</td><td>&lt;4.9 mmol/L;</td><td>consequences;</td></lin> | <6.2 - 4.9 mmol/L; | <4.9 mmol/L; | consequences; |
| or g/L) | | mmol/L; | <100 - 80g/L | <80 g/L; | |
| | | <lln -100="" g="" l<="" td=""><td></td><td></td><td></td></lln> | | | |
| Platelet (/mm3 or | <b>→</b> | - CLIN - | <75,000 - | <50,000 - | <25,000/mm3; |
| (L) | | 75,000/mm3; | 50,000/mm3; <75.0 | 50,000/mm3; <75.0 25,000/mm3; <50.0 <25.0 x 10e9 /L | <25.0 x 10e9 /L |
| | | <lln -="" -50.0="" 10e9="" 75.0="" l<="" td="" x="" =""><td>-50.0 x 10e9 /L</td><td>- 25.0 x 10e9 /L</td><td></td></lln> | -50.0 x 10e9 /L | - 25.0 x 10e9 /L | |
| | | /L | | | |
| Neutrophils (/mm3 | <b>→</b> | <lln -="" 1500="" mm3;<="" td=""><td><pre><lln -="" 1000="" 1500="" 500="" <1000="" <1500="" mm3;="" mm3;<="" pre="" =""></lln></pre></td><td>&lt;1000 - 500/mm3;</td><td>&lt;500/mm3; &lt;0.5 x</td></lln> | <pre><lln -="" 1000="" 1500="" 500="" <1000="" <1500="" mm3;="" mm3;<="" pre="" =""></lln></pre> | <1000 - 500/mm3; | <500/mm3; <0.5 x |
| or /L) | | <lln -="" 1.5="" l="" p="" x109="" <=""></lln> | <lln -="" 0.5="" 1.0="" 1.5="" <1.0="" <1.5="" l="" l<="" p="" x109="" x10e9="" =""></lln> | | 10e9 /L |
| Lymphocyte (/mm3 | | <lln -="" 800="" mm3;<="" td=""><td>&lt;800 - 500/mm3;</td><td>&lt;500 - 200/mm3;</td><td>&lt;200/mm3;</td></lln> | <800 - 500/mm3; | <500 - 200/mm3; | <200/mm3; |
| or /L) | | <lln -="" 0.5="" 0.8="" <0.8="" l<="" td="" x10e9="" =""><td>&lt;0.8 - 0.5 x10e9 /L</td><td>&lt;0.5 - 0.2 x10e9 /L</td><td>&lt;0.2 x 10e9 /L</td></lln> | <0.8 - 0.5 x10e9 /L | <0.5 - 0.2 x10e9 /L | <0.2 x 10e9 /L |
| | | /L | | | |
| Note: $10e9 = 10^9$ : L.I.N = L.ov | N = Lower Limit of N | wer Limit of Normal: ULN = Upper Limit of Normal | imit of Normal | | |

CONFIDENTIAL TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Symphogen A/S Sym015-01

Statistical Analysis Plan

# 7.2 Derivation of CTCAE Grade - Clinical Chemistry Tests

| Tests | Direction | | Gr | Grade | |
|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 |
| Sodium (mmol/L) | $\rightarrow$ | <lln -="" 130<br="">mmol/L</lln> | • | <130 - 120 mmol/L | <120 mmol/L |
| Sodium (mmol/L) | <b></b> | - 150 | >150 - 155 mmol/L | >155 - 160 mmol/L | >160 mmol/L |
| Potassium<br>(mmol/L) | $\rightarrow$ | <lln -="" 3.0="" l<="" mmol="" td=""><td>•</td><td>&lt;3.0 - 2.5 mmol/L</td><td>&lt;2.5 mmol/L</td></lln> | • | <3.0 - 2.5 mmol/L | <2.5 mmol/L |
| Potassium<br>(mmol/L) | <b>←</b> | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >5.5 - 6.0 mmol/L | >7.0 mmol/L |
| Glucose | <b>→</b> | <lln -="" 55="" dl;<br="" mg=""><lln -="" 3.0="" l<="" mmol="" td=""><td>&lt;55 - 40 mg/dL;<br/>&lt;3.0 - 2.2 mmol/L</td><td>&lt;40 - 30 mg/dL;<br/>&lt;2.2 - 1.7 mmol/L</td><td>&lt;30 mg/dL;<br/>&lt;1.7 mmol/L</td></lln></lln> | <55 - 40 mg/dL;<br><3.0 - 2.2 mmol/L | <40 - 30 mg/dL;<br><2.2 - 1.7 mmol/L | <30 mg/dL;<br><1.7 mmol/L |
| Glucose | ← | Fasting glucose value > ULN - | Fasting glucose value > 160 - | >250 - 500 mg/dL;<br>>13.9 - 27.8mmol/L | >500 mg/dL;<br>>27.8 mmol/L |
| | | 160 mg/dL; | 250 mg/dL; | | |
| | | Fasting glucose | Fasting glucose | | |
| | | value >ULN - 8.9 | value >8.9 - 13.9 | | |
| | | mmol/L | mmol/L | | |
| Creatinine | <b>↓</b> | >1 - 1.5 x baseline; | >1.5 - 3.0 x | >3.0 baseline; | >6.0 x ULN |
| | | >ULN - 1.5 x ULN | baseline; | >3.0 - 6.0 x ULN | |
| Bilimbin | <b>←</b> | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN |
| Alkaline | ← ← | | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| phosphatase (AKP) | | | | | |
| AST (SGOT) | <b>↓</b> | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| ALT (SGPT) | <b>+</b> | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Uric Acid | <b>←</b> | >ULN - 10 mg/dL | | * | >10 mg/dL;<br>>0.59 mmol/L |
| | | (0.39 IIIII01/L) | | | |

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Symphogen A/S Sym015-01

Statistical Analysis Plan

| Tests | Direction | | Gr | Grade | |
|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 |
| Calcium | ← | Corrected serum | Corrected serum | Corrected serum | Corrected serum |
| | | calcium of | calcium of | calcium of | calcium of |
| | | Hypercalcemia | >11.5 - 12.5 mg/dL; | >12.5 - 13.5 mg/dL; | >13.5 mg/dL; |
| | | >ULN - 11.5 | 11.5 >2.9 - 3.1mmol/L; | >3.1 - 3.4 mmol/L; | >3.4 mmol/L; |
| | | mg/dL; | Ionized calcium | Ionized calcium | Ionized calcium |
| | | >ULN - 2.9 | 2.9 >1.5 -1.6 mmol/L | >1.6 - 1.8 mmol/L | >1.8 mmol/L |
| | | mmol/L; | | | |
| | | Ionized calcium | | | |
| | | >ULN - 1.5 mmol/L | | | |
| Calcium | $\rightarrow$ | Corrected serum | Corrected serum | Corrected serum | Corrected serum |
| | | calcium of | calcium of | calcium of | calcium of |
| | | <lln -="" 8.0="" dl;<="" mg="" td=""><td>&lt;8.0 - 7.0 mg/dL;</td><td>&lt;8.0 - 7.0 mg/dL;</td><td>&lt;6.0 mg/dL;</td></lln> | <8.0 - 7.0 mg/dL; | <8.0 - 7.0 mg/dL; | <6.0 mg/dL; |
| | | <lln -="" 2.0<="" td=""><td>2.0 &lt;2.0 - 1.75 mmol/L;</td><td>&lt;2.0 - 1.75 mmol/L;</td><td>&lt;1.5 mmol/L;</td></lln> | 2.0 <2.0 - 1.75 mmol/L; | <2.0 - 1.75 mmol/L; | <1.5 mmol/L; |
| | | mmol/L; | Ionized calcium | Ionized calcium | Ionized calcium |
| | | Ionized calcium | <1.0 - 0.9 mmol/L; | <1.0 - 0.9 mmol/L; | <0.8 mmol/L; |
| | | <lln< td=""><td></td><td></td><td></td></lln<> | | | |
| | | -1.0 mmol/L | | | |
| Phosphate | $\rightarrow$ | <lln -="" 2.5="" dl;<="" mg="" td=""><td>&lt;2.5 - 2.0 mg/dL;</td><td>&lt;2.0 - 1.0 mg/dL;</td><td>&lt;1.0 mg/dL;</td></lln> | <2.5 - 2.0 mg/dL; | <2.0 - 1.0 mg/dL; | <1.0 mg/dL; |
| | | <lln -="" 0.6="" 0.8="" <0.8="" l="" l<="" mmol="" td="" =""><td>&lt;0.8 - 0.6 mmol/L</td><td>&lt;0.6 - 0.3 mmol/L</td><td>&lt;0.3 mmol/L</td></lln> | <0.8 - 0.6 mmol/L | <0.6 - 0.3 mmol/L | <0.3 mmol/L |
| Note: $10e9 = 10^9$ ; <b>LL</b> | N = Lower Limit of N | Note: 10e9 = 10 <sup>9</sup> ; LLN = Lower Limit of Normal; ULN = Upper Limit of Normal | imit of Normal | | |

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

Symphogen A/S Sym015-01

Statistical Analysis Plan

# 7.3 Derivation of CTCAE Grade - Coagulation Tests

| Tests | Direction | | G | Grade | |
|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 |
| Activated partial | <b>←</b> | >ULN - 1.5 x ULN >1.5 - 2.5 x ULN | $>1.5 - 2.5 \times ULN$ | >2.5 x ULN; | |
| thromboplastin time | | | | hemorrhage | |
| prolonged | | | | | |
| Fibrinogen | <b></b> | <1.0 - 0.75 x LLN | <0.75 - 0.5 x LLN | <1.0 - 0.75 x LLN <0.75 - 0.5 x LLN <0.5 - 0.25 x LLN <0.25 x LLN or | <0.25 x LLN or |
| decreased | | or <25% decrease | or 25 - <50% | or 50 - <75% | 75% decrease from |
| | | from baseline | decrease from | decrease from | baseline or absolute |
| | | | baseline | baseline | value <50 mg/dL |


TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019

Symphogen A/S Sym015-01

Statistical Analysis Plan

## Schedule of Assessments - Part 1 and Part 2 Basket Cohort 7.4

| Pre-Trestment Period | | | | | | Ē | Trestment Period | Tried, | | | | Post-Trest | Post-Trestment:Periog? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | Cycle 1 | | | 8 | Cycle 2, 4, 6 etc. | 6 ekc. | Pý | Cyde 3, 5, 7 | EOT | 1M FUP |
| Day wethin Cycle<br>Viet Window (= day). | D-14 to D-1 | řá. | ä | 2 <u>7</u> | 015<br>(=3) | 88<br>8 | ម្ចីភ | 510<br>E=1 | End of<br>Cycle | កឃឹ | (년)<br>(년) | 10 d iollowing the decision of this treatment | Spout after last<br>dose of mal<br>readment<br>(30—70) |
| Informed Conseni | 54 | | | | | | | | | | | | |
| Baseline Changements Elimbility | × | × | | | | | | | | | | | |
| Safety Assessments | | | | | | | | | | | | | |
| Medicanon-Procedure Survey | × | × | | | × | | 24 | >: | | × | 14 | и | H |
| (S)AE Survey and Personing | k | برز | برز | И | × | × | × | и | × | × | j-4 | и | × |
| CLT Evaluation.<br>Part 1/Dose-Escalation only | | × | × | ы | и | × | C) entr | | | | | | |
| Viral Signs and Body Weight | × | × | | | × | | :4 | بسز | | × | بسرا | 1 | X |
| ECOG 35* | 14 | S: | | | | | × | | | H | | × | X |
| Physical Examination? | и | × | | Γ | | | × | | | M | | × | × |
| ECG | × | | | | | | | | | | | н | |
| ECHO or MUCA scan? | M | | | | | | | | | | | | |
| Safery blood samples** | и | بر: | × | × | × | × | ы | × | | ы | ы | 1 | X |
| Unimakens | м | 'n | | | H | | × | | | iv; | | × | X |
| Premancy Test | и | | | | | | | | | | | × | |
| Disease Assessments | | | | 1 | | | | | | | | | |
| Disease Status Evabanou by CT MR? | и | | | | | | | | X | | | X). | ,X |
| Turnot Marker Evaluation" | × | | | | | | | | Х | | | × | × |
| Archival Tursor Tissue (may include pre-<br>screening by liquid (x))? | X | | | | | | | | | | | | |
| Turker Biopsy <sup>13</sup> | X | | | | | | | | C. only'' | | | | |
| Additional Assessments | | | | 1 | | | | | | | | | |
| P.F. Samples <sup>1</sup> 1 | | × | بر: | M | × | | بسا | <u>بر</u> | | и | × | × | × |
| ADA Sanye'' | | и | | | | | on's | | | × | | ы | × |
| Skin Bropsy <sup>44</sup><br>Part L'Dose-Escabation only | X | | | | | | | | C2 enh <sup>3</sup> : | | | | |
| Biomerker Blood Sample! | × | | | | | | | | Cl only | | | × | |
| Trial Treatment | | | | | | | | | | | | | |
| Symflij Premeditatsko" | | بسز | | | × | | j | М | | يبز | 14 | | |
| Sym035 Prinsion | | × | | | × | | × | 1 | | × | × | | |
| Post-itrasion Monitoring | | И | | | и | | H | i-4 | | × | 4 | | |

TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Symphogen A/S Sym015-01

### Statistical Analysis Plan

Abbreviations (m. alphabetical order), ADA, ann-thra mifoddy, Bv. biopay, C. Cycle, U.T. computed knowangapty scan, D.A. days, D.L.T. days-business control. End of Treament Vierr. EU.G. alexandratic extraorationatic (2007), every second needs, (3).4E. (senous) interest event. T.X. therapy

- The treatment period condusts until the patient is withdrawn from 3 yal015
- After the IM FIP Visit, the investigator will make every effort to chaim follow-up information on response assestment of consent, and the IM FUP Visit and PD or another theopetic intervention is included follow-up is required uncl death, middlewal of consent, and it is experted to the consent of consent, and it is experted of the consent of the consent follow-up does not require at the person visit in the trial site, but may be obtained by collection of date focus and another does not require at the person visit in the trial site, but may be obtained by collection of date focus and another date of the consented follow-up does not require at the person visit in the trial site, but may be obtained by collection of date focus and the consented by the consented follow-up does not require the trial site, but may be obtained by collection of date for the consented follow-up does not require the trial site, but may be obtained by collection of date for the consented follow-up does not require the consented for t
  - Screening assessment unlude demographes, medical bistory, rumot bistology, nutradon starus, extent of disease, prior aon-causer neemvant, etc 海辛
- DLT evaduation, applicable for Part House escalation cohorts and OLIs we reponed during Cycke I with 2 fami assessment if (e.) days after the last dose of Cycle I or prior to dosing on
- Does not cased to be parformed prior to C LET if parformed during screening  $_{-}$   $^{\circ}$  days from CL DL
- In addition to the acheduled consporat, on ECHONCGA should be performed in the event of cardon symptoms and as otherwise abuscally indicoted In addition to the scheduled temporitie, an ECG should be performed if clearcally indicated a or a a
  - Local laboratory results must be available and assessed prior to each SpacO3 infusion. Refer to Section 5.2 9 for denails
- T or MNI subgrag schedule and conditions, applying to all cohoras:
- A CTMR performed within 28 days prior to CFD can be used for evaluation of eligibility and as baseline scan provided that the CTMR has been performed according to the priority
- The first CTAR2 assessment for response ts doze at the and of Cycle 2 and thereaffer repeated at the end of every second cycle (in the week prior to Day L of the next cycle)
  - In the event of suspected PD, a CTMRI is to be performed as soon as possible.
- In the even of CRPR, a confirmancy CTMPL is to be performed to earlier than 13 days after the first assessment of CRPR.
- A CTMM at DOL should ach, be performed that previous CTMM has been performed as weaks before A CTMM som at IMFOs should only be performed that CTMM documents ID ŝ
- 11). Twencreaker evoluanen to meinde tumor markers that are pan of the trud site streedand practices as indicated by rumer 150 if applicable
- Archival rumor resue. To be assessed locally. Does not need to be repeneed if AEE sumplification and AEAs: musticially arrange been assessed precreasily and the publicing report is available to For Part 2-Basket Colont. In preferred that the local eligibility arrestment for M.F-angulations will be done unit that a form a finish burse, consented that the integration of architectual fiscue is not available, these a four a finish performed during screeming will be used. Periphent blood collection for MACF-angulation assessment and for MEF-angulation assessment as called the figure broggy) is allowed as a local pre-screening methodology by Grandhalbly makes. Other liquid budgiy 2
- For Part 2-Backet Cobort: Required, to be assessed cumuly. Tistue from a rango bages, performed during streeting is predicted, however archival rasses may be arbitrated from the forestation of dispersion, provided the archival casine is numble for central analysis for central analysis to be repeated at the end of Cycle I or upon PO. whichever occurs first. Tamov Nopyr. To de 22sessed iscally as pair of elegivitiv. 28seanoer in Zard 2 and Pard 2, if agolicable Optional for patients with known MET-amplification encolled in Part 1 For Part 2-NSCLC Cohorn Archival nasae to be submitted, if available Refer to Section 3.3 4 for details m

methodologies, except if used to detect *NETe*st!+ munadon, will ouly be adlowed if previously approved by the Spousor

- For Part 2-NSCLC Cohorn: Biograms are openand in the narrooms specified
  - Entended PK sampling for  $\overline{\rm PK}$  profiling will be done remarg (1.10) . Refer to Table 2 for details
    - Only applicable for Part 2: ADA sample on first day of Cycle 2, prior to desing
- Oaly applicable for Part 1. Skin biogsy is obtained clima screezing after gainem eligibility has been confirmed Sampling is repeated in the end of Cycle 1 or upon PD, whichever occurs first
- Biomarker blood sample is taken during streeting after pattern eligibility has been confirmed. Sampling is repeated at the end of Cycle I or upon PD, whichever occurs first, and st EOI. If a remort blood sample, the biomarker blood sample should be collected after to collecting the rimor blogsy.
  - For Part I of the mial premedication is manchonery prior to each dose of Symblic For Part 2 of the mial premedication is manchonery prior to each dose of Symblic Circle I La Part 2. premedication may be withfurwn after Cycle 1 on a gather-by-parkent base if the content evidence evidence related restructs. Refer to Section 11 for details


Symphogen A/S Sym015-01

Statistical Analysis Plan

## Schedule of Assessments - Part 2 NSCLC Cohort 7.5

| Pro-Treatment Period | | | | | | A | Trestment Period | eriod, | | | | Post-Treats | Post-Treatment Period <sup>1</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | 1 | ľ | Cycle 1 | | T | 5 | Crcle 3, 4, 6 etc. | 6 etc. | Cycle 3, | Cycle 3, 5, 7 etc. | EOT | 1M FUP |
| Day within Cycle<br>Vise Wradow (= days) | 3-14 te D-1 | E | 23 | គ <u>ី</u> | 10<br>E3 | (=) | <b>高</b> | E € | 30g | [년] | D25<br>(=2) | 1.C d following the decision of trial treatment trialdrawal | ] month after just<br>dosa of trial<br>rearment<br>(3C-74) |
| Teformed Consent | х | | | | | | | | | | | | |
| Baseline Characteristics Elembistry | 7. | и | r | | Ī | İ | | | | | | | |
| Safety Assessments | | | | | | | | | | | | | |
| Medicanco Procedure Survey | × | × | | | × | Г | И | M | | <b>!</b> ! | <b>&gt;</b> : | × | и |
| (SLAE Survey and Reparting | × | × | × | × | и | × | × | и | Х | × | × | × | и |
| Viral Signs and Body Weight | × | <b>&gt;</b> 4 | | | и | | 7 | И | | × | × | х | и |
| E006.PS+ | × | Ř | Г | | | | × | | | X | | × | × |
| Physical Examination* | × | 1,1 | | | | | Х | | | × | | × | × |
| ECC. | ۵: | | | | | | | | | | | ы | |
| ECHO or MUGA son: | × | | | | | | | | | | | | |
| Safety blood samples | и | 'n | × | × | × | × | 4 | H | | بسنة | <b>;</b> 4 | برز | М |
| Uncakeis** | æ | ě | | | × | | × | | | H | | и | jur; |
| Dregmany Ter | и | | | | | | | | | | | × | |
| Disease Assessments | Service Services | | | | | | | | | 200 | | | |
| Disease Status Evaluation by CLMRT | Х | | H | H | H | П | | | х | | | × | × |
| Tunor Bionsy* | х | | | | | | | | EOC : ouiv | | | | |
| Additional Assessment: | | | 10 | | | | | | | | | | |
| PK Samples⁺ | | × | × | ĸ | × | | ы | И | | × | × | <b>&gt;</b> : | М |
| ADA Sample | | پر: | | | | | ी श्वार | | | إمرا | | × | بسز |
| Genomic Biomarker Blood Sample! | × | | Н | | | | | | EUC. oain | | | × | |
| Trial Treatment | | | | | 272 | | | | | | | | The State of Lines. |
| Sampli Framedicanon; | | <u>-</u> | | | × | | <b>:</b> 4 | :4 | | بر: | <b>1</b> 4 | | |
| Symyle Hefusion | | × | | | × | | × | и | | × | × | | |
| Jose-Tráisien Montiona | | :4 | | | и | | j, orț | × | | X | × | | |

CONFIDENTIAL TP-GDO-WW-133-01 Effective Date: 05 Sep 18 Related to: SOP-GDO-WW-019


Abbreviator, in alpubenci celet. ADA metary ambode, By, hoper C. Ciele CI compared lonography scan D.4. drys. DLT dose luming south. EOC. End of Cycle. EOI. End of EoI. End of Cycle. EOI. End of Cycle. End of Cycle. EOI. End of Cycle.

Iteament Penos). The Deancear period communes until the panear is withfrawn from Sym21.5

Post-framest Penol. After the IN FLP Vist. the investigator will make every effor to obtain follow-up information on response sisteriness and or OS about once every 1 mouths. Personse sisteriness and or OS about once every 1 mouths. Personse sisteriness and of about 1 million on the IN FLP Vist. will for include the appears increased for million of the information and of the information of

Baieline (Janaciensico Chabilin). Screening assessments sicidde denographica, medical bistori, rumot distology, mungon sants, event of diesse, pate announces mestment est

ECO. In addition to the scheduled amegodish, in ECO inould be performed if chancilly indicated

ECHOMIGA in addition to the scheduled timepoint, at ECHOMIGA though be performed in the event of cardiac symptoms and 35 otherwise clinically indicated Blood sulen Samoles Cranshing. Lotal abbrancoy results must be available and assessed prost to each Symbly inclusion. Refer to Section 3.1.9 for details Distre Sons Evglusion (T et MP2 unspag schedule and condinger.

A CT ME. performed within 18 days prior to C1 D1 can be used for evaluation of eligiblish and as baseline scar, provided that the CT M21 has been performed according to the prooted The first CTARL stressment for response to foce at the EOCO and thereafter repeated at the end of every second cycle (EOC) assessment may be performed at any time during the weak process of the new cycle, including Day 1 of the new cycle prior to forting provided tendin are available growth that examinimation;

in the event of CR. PR. 2 confirmatory CT MRI is to be performed to eather than 18 days taker the first attestment of CR. PR

ō.

ACTME at EQT goods only be pariorised if the previous CTMELkin bear parformed. I weeks before ACTMELican at IMFUP should only be performed if no CTME, documents 9

Tuner Boden or newly performed tropies are mandatory at creetury, it is permissible to perform the presenting procedure outside the 14-day screening penod provided informed conservables outside the 14-day screening penod provided informed conservables of the conserv Seconic Bonaria et Blood Sample. It is permissible to obtain the stateming sample outside the 1-thy streeming period provided informed consent for the wall has been obtained. Subsequent of a sample to be obtained upon 20. If a namer keopity is collected at the same time point is the bonaries. No bonaries blood sample the bonaries blood sample inconfined from collected at the same time point is the bonaries blood sample inconfid be collected at the same time point is the bonaries blood sample inconfid be collected after the collected at the same time point is the bonaries blood sample inconfid be collected at the same time point is the bonaries blood sample inconfid be collected after the collected at the same time point is the bonaries.

û

Planedication Munchoop part to each tone of Symble during Cycle L may be carbidrann after Cycle L on a patient-by-panen bases if the patient is nations eardence of influsion relared

CONFIDENTIAL Related to: SOP-GDO-WW-019 Effective Date: 05 Sep 18 TP-GDO-WW-133-01


Document ID: 516730473 - Name at Publication: 223276 SAP 20190605 V 1 0.pdf This document contains a total of 86 pages including any signature page/s.

### Electronic Signature Page

This page is the manifestation of the electronic signature(s) used in compliance with International's electronic signature policies and procedures and in compliance with applicable regulations.

UserName

Title: Senior Biostatistician, GDO

Date: Friday, 21 June 2019, 02:07 PM GMT Standard Time

Meaning: Document contents approved.